

#### CLINICAL STUDY PROTOCOL

Study Title: A Phase 2, Double-Blind, Randomized Study Evaluating the

Safety, Tolerability, and Efficacy of GS-4997 in Combination with Prednisolone versus Prednisolone Alone in Subjects with Severe

Alcoholic Hepatitis (AH)

Sponsor: Gilead Sciences, Inc.

**IND Number**: 129570

**EudraCT Number:** 2016-000821-37

Clinical Trials.gov

Identifier: NCT02854631

Indication: Alcoholic Hepatitis (AH)

Protocol ID: GS-US-416-2124

Gilead Medical Monitor: Name: Chuhan Chung, MD

Telephone: PPD

Fax: PPD Email: PPD

Protocol Version/Date: Original: 12 April 2016

Amendment 1: 02 June 2016 Amendment 2: 11 January 2017 Amendment 3: 04 August 2017

#### CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| TAE | BLE O | CONTENT | S | 2 |
|---|---|---|---|---|
| LIST | Γ OF I | N-TEXT TAE | BLES | |
| LIST | Г ОБ П | N-TEXT FIG | URES | 4 |
| PRO | TOCC | L SYNOPSI | S | $\epsilon$ |
| | | | EVIATIONS AND DEFINITION OF TERMS | |
| 1. | INTR | | | |
| | 1.1. | Background | | |
| | 1.2. | | General Information | |
| | | | Preclinical Pharmacology and Toxicology | |
| | | | Clinical Trials of GS-4997 | |
| | | | A Phase 2, Double-blind, Placebo-controlled, Dose-ranging Study | , |
| | | | Evaluating the Efficacy, Safety, and Tolerability of GS-4997 in Subjects | |
| | | | with Diabetic Kidney Disease (Study GS-US-223-1015) | 26 |
| | | 1.2.5. | A Phase 2, Dose-ranging, Randomized, Double-blind, Placebo-controlled | 2( |
| | | 1.2.3. | Study of GS-4997 in Subjects with Pulmonary Arterial Hypertension | |
| | | | (Study GS-US-357-1394) | 27 |
| | | 1.2.6. | A Phase 2, Randomized, Open Label Study Evaluating the Safety, | |
| | | | Tolerability, and Efficacy of GS-4997 alone or in Combination with | |
| | | | Simtuzumab (SIM) in Subjects with Nonalcoholic Steatohepatitis | |
| | | | (NASH) and Fibrosis (F2-F3) (GS-US-384-1497) | 28 |
| | 1.3. | | For This Study | |
| | 1.4. | | For Dose Selection | |
| | 1.5. | | fit Assessment for the Study | |
| | 1.6. | | e | |
| 2. | OBJE | CTIVES | | 32 |
| 3. | STUI | Y DESIGN. | | 34 |
| | 3.1.<br>3.2. | | gnPlan and Regimen | |
| | 3.2. | | Testing Testing | |
| | 3.3. | | Biomarker Samples to Address the Study Objectives | |
| | | | Biomarker Samples for Optional Future Research | |
| | | | Biomarker Samples for Optional Genomic Research | |
| 4 | CLIDI | | | |
| 4. | SUBJECT POPULATION | | | 40 |
| | 4.1. | | Subjects and Subject Selection | |
| | 4.2. | | Criteria | |
| | 4.3. | Exclusion | Criteria | 41 |
| 5. | INVE | STIGATION | AL AND NON-INVESTIGATIONAL MEDICINAL PRODUCTS | 44 |
| | 5.1. Randomization, Blinding and Treatment Codes | | 44 | |
| | | | Procedures for Breaking Treatment Codes. | |
| | 5.2. | | n and Handling of Study Drugs | |
| | | | Formulation | |
| | | 5.2.2. | Packaging and Labeling | 45 |
| | | | Storage and Handling | |
| | 5.3. | Dosage and | d Administration of Study Drugs | 46 |

| | 5.4.<br>5.5. | 5.3.1. GS-4997 5.3.2. Prednisolone Prior and Concomitant Medications Prohibited Medications | 46<br>46 |
|---|---|---|---|
| | 5.6. | Study Drug Accountability | |
| 6. | STUE | DY PROCEDURES | |
| | 6.1. | | |
| | 6.2. | Pretreatment Assessments | |
| | | 6.2.1. Screening Visit | 49 |
| | | 6.2.2. Baseline / Day 1 Assessments and Randomization | |
| | 6.3. | Treatment Assessments | |
| | | 6.3.1. Week 1 Visit (±3 Days) | |
| | | 6.3.2. Week 2 Visit (±3 Days) | |
| | | 6.3.3. Week 3 Visit (±3 Days) | |
| | | 6.3.4. Week 4 / End of Treatment Visit (EoT) (±3 days) | |
| | 6.4. | 6.3.5. Follow Up Visit (±5 Days) | |
| | 0.4. | 6.4.1. Sparse PK | |
| | | 6.4.2. Intensive PK Substudy | |
| | 6.5. | Post-Treatment Assessments | |
| | 0.5. | 6.5.1. Week 6 (± 3 Days) | |
| | | 6.5.2. Weeks 8, 16, and 20 / Post Treatment Visits (± 5 Days) | |
| | | 6.5.3. Weeks 12 and 24 / Post Treatment Visits (± 5 Days) | |
| | 6.6. | . Unscheduled Visits | |
| | 6.7. | Assessments for Premature Discontinuation from Study | |
| | 6.8. | Criteria for Discontinuation of Study Treatment. | |
| | 6.9. | Description of Assessments | |
| | | 6.9.1. Liver Biopsy | |
| | | 6.9.2. Electrocardiogram | |
| | | 6.9.3. AUDIT / SADQ Questionnaires | |
| | | 6.9.4. Quality of Life (QoL) Measures | |
| | | 6.9.5. Hepatic Encephalopathy (HE) | |
| | | 6.9.7. Maddrey's DF, MELD and Child-Pugh-Turcotte Scores | |
| | | 6.9.8. Hepatorenal Syndrome (HRS) | |
| | | 6.9.9. Infection | |
| | | 6.9.10. Screening Laboratory Assessments | |
| | | 6.9.11. FibroScan® | |
| | | 6.9.12. Lille Score | |
| | 6.10. | End of Study Definition | |
| 7. | ADVI | ERSE EVENTS AND TOXICITY MANAGEMENT | 71 |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | 71 |
| | | 7.1.1. Adverse Events | |
| | | 7.1.2. Serious Adverse Events | 71 |
| | | 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as | |
| | | Adverse Events or Serious Adverse Events | |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | | 7.2.2. Assessment of Severity | 73 |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | 72 |
| | | Adverse Events to Gilead | |

| | 7.4.<br>7.5. | Gilead Reporting Requirements Toxicity Management | |
|---|---|---|---|
| | | 7.5.1. Assessment of Potential Drug-Induced Liver Injury by an Independent Adjudicator | |
| | 7.6. | Special Situations Reports. | |
| | | 7.6.1. Definitions of Special Situations | 77 |
| | | 7.6.2. Instructions for Reporting Special Situations | 78 |
| 8. | STAT | TISTICAL CONSIDERATIONS | 80 |
| | 8.1. | Analysis Objectives and Endpoints | |
| | | 8.1.1. Primary Endpoint | |
| | 8.2. | Secondary Endpoints | |
| | | 8.2.1. Exploratory Endpoints | |
| | 8.3. | Analysis Conventions | |
| | | 8.3.1. Analysis Sets | |
| | 8.4. | Data Handling Conventions | |
| | 8.5. | Demographic Data and Baseline Characteristics | |
| | 8.6. | Primary Analysis | |
| | 8.7. | Efficacy Analysis | |
| | 0.0 | 8.7.1. Exploratory Analysis | |
| | 8.8. | Safety Analysis | |
| | | 8.8.1. Extent of Exposure 8.8.2. Adverse Events | |
| | | 8.8.3. Laboratory Evaluations | |
| | | 8.8.4. Other Safety Evaluations | |
| | 8.9. | Pharmacokinetic Analysis | |
| | 0.9. | 8.9.1. Other Exploratory Analyses | |
| | 8.10. | Sample Size | |
| | 8.11. | Data Monitoring Committee | |
| 9. | RESP | PONSIBILITIES | 87 |
| | 9.1. | Investigator Responsibilities | 87 |
| | | 9.1.1. Good Clinical Practice | |
| | | 9.1.2. Institutional Review Board (IRB)/Independent Ethics Committee | |
| | | (IEC)/Ethics Committee (EC) Review and Approval | 87 |
| | | 9.1.3. Informed Consent | |
| | | 9.1.4. Confidentiality | |
| | | 9.1.5. Study Files and Retention of Records | |
| | | 9.1.6. Electronic Case Report Forms | |
| | | 9.1.7. Investigational Medicinal Product Accountability and Return | |
| | | 9.1.8. Inspections | |
| | | 9.1.9. Protocol Compliance | |
| | 9.2. | Sponsor Responsibilities | |
| | | 9.2.1. Protocol Modifications | |
| | 0.2 | 9.2.2. Study Report and Publications | |
| | 9.3. | Joint Investigator/Sponsor Responsibilities | |
| | | 9.3.1. Payment Reporting | |
| | | $oldsymbol{arepsilon}$ | |
| | | <ul><li>9.3.3. Monitoring and Oversight of Biomarker Specimens</li><li>9.3.4. Access to Information for Auditing or Inspections</li></ul> | |
| | | 9.3.5. Study Discontinuation | |
| 10. | REFE | ERENCES | |
| 11. | | ENDICES | |
| | | | · |

| Appendix 1. Appendix 2. | Investigator Signature Page Study Procedures Table | 98<br>99 |
|---|---|---|
| Appendix 3. | Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements. | |
| Appendix 4. | Child-Pugh-Turcotte (CPT) Classification of the severity of cirrhosis | |
| | LIST OF IN-TEXT TABLES | |
| Table 3-1. | Biomarkers | 36 |
| Table 5-1. | | |
| | LIST OF IN-TEXT FIGURES | |
| Figure 3-1 | Overall Study Design | 34 |

# **PROTOCOL SYNOPSIS**

Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404

| Study Title: | A Phase 2, Double-Blind, Randomized Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 in Combination with Prednisolone versus Prednisolone Alone in Subjects with Severe Alcoholic Hepatitis (AH) |
|---|---|
| IND Number: EudraCT Number: Clinical Trials.gov Identifier: | 129570<br>2016-000821-37<br>NCT02854631 |
| identifier: | NC102834031 |
| <b>Study Centers Planned:</b> | Multiple centers in North America and Europe |
| Number of Subjects<br>Planned: | Up to 120 subjects will be randomized in order to obtain 100 subjects with biopsy-proven severe AH |
| Target Population: | Males and non-pregnant, non-lactating females between 18-70 years of age with histologically-confirmed severe alcoholic hepatitis (Maddrey's Discriminant Function [Maddrey's DF] ≥ 32). |
| Duration of Study: | Participation in the study can last up to 26 weeks, which includes a 2-week Screening period, a 4-week treatment period, and a 20-week post treatment period. |
| Objectives: | The primary objective of this study is as follows: |
| | To evaluate the safety and tolerability of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe AH. |
| | The secondary objectives of this study are as follows: |
| | • To assess changes in hepatic synthetic function [liver biochemistry, Model for End-Stage Liver Disease [MELD] score, Child-Pugh score, the Lille model, and Maddrey's Discriminant Function (Maddrey's DF)]; |

- To assess mortality at 28 days, 8 weeks, 12 weeks, and 24 weeks;
- To determine the incidence of liver transplantation;
- To determine the incidence of hepatorenal syndrome (HRS);
- To determine the incidence of infection;
- To assess length of hospital stay.

The exploratory objectives of this study are:



#### **Study Design:**

This is a Phase 2, double blind, proof-of-concept, randomized study evaluating the safety, tolerability, and biological activity of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe, histologically-confirmed AH.

Up to 120 subjects (for 100 evaluable AH subjects) will be randomized within strata (1:1) to either:

1. Group A (n = 50-60):

GS-4997 18 mg once daily + prednisolone 40 mg once daily for 28 days

OR

2. Group B (n = 50-60):

GS-4997 placebo once daily + prednisolone 40 mg once daily for 28 days

Randomization will be stratified by MELD  $\leq$  or  $\geq$  25 at Screening (based on local laboratory testing).

To allow for diagnoses inconsistent with severe AH in up to 20% of subjects based on liver biopsy findings, we will target randomization of up to 120 subjects into the study.

# Diagnosis and Main Eligibility Criteria:

#### **Inclusion Criteria:**

- 1) Males and non-pregnant, non-lactating females between 18-70 years of age, inclusive based on the date of the Screening visit;
- 2) Willing and able to give informed consent prior to any study specific procedures being performed. In subjects with hepatic encephalopathy (HE) which may impair decision-making, consent will be obtained per hospital procedures (eg, by Legally Authorized Representative);
- 3) Clinical diagnosis of severe AH based on all of the following:
  - a) History of excessive alcohol consumption during the past 3 months (average of > 40 g/d of alcohol for women and > 50 g/d for men);
  - b) Aspartate aminotransferase (AST) ≥ 50 U/L, based on local laboratory results;
  - c) AST/alanine aminotransferase (ALT) ratio (AST/ALT) ≥ 1.5, based on local laboratory results;
  - d) Onset of jaundice within the past 3 months;
  - e) Maddrey's DF  $\geq$  32 at Screening, based on local laboratory results;

- 4) All female subjects of childbearing potential must agree to use a highly effective method of contraception during intercourse from the Screening visit throughout the study period and for 90 days following the last dose of study drug. If females utilize hormonal agents as one of their contraceptive methods, the same hormonal methods must have been used for at least 3 months before study dosing. Females on hormonal methods must also utilize a barrier method as another form of contraception as described in Appendix 3;
- 5) Male subjects must agree to use condoms during intercourse from Screening through study completion and for 90 days following the last dose of study drug;
- 6) Male subjects must refrain from sperm donation from Screening through at least 90 days following the last dose of study drug;
- 7) Female subjects must refrain from egg donation or harvest for 90 days after last dose of study drug;
- 8) Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.

# **Exclusion Criteria:**

- 1) Pregnant or lactating females;
- 2) Other causes of liver disease including chronic hepatitis B (hepatitis B surface antigen [HBsAg] positive), chronic hepatitis C (HCV RNA positive), acetaminophen hepatotoxicity, biliary obstruction, and autoimmune liver disease;
- 3) Serum AST > 400 U/L or ALT > 300 U/L, based on local laboratory results;
- 4) MELD > 30 at Screening, based on local laboratory results;
- 5) Maddrey's DF > 60 at Screening, based on local laboratory results;
- 6) Grade 4 HE by West Haven criteria;
- 7) Concomitant or previous history of hepatocellular carcinoma;
- 8) History of liver transplantation;
- 9) HIV Ab positive;
- 10) Clinical suspicion of pneumonia;

- 11) Uncontrolled sepsis;
- 12) Uncontrolled gastrointestinal (GI) bleeding or controlled GI bleeding within 7 days of Screening that was associated with shock or required transfusion of more than 3 units of blood;
- 13) Type 1 hepatorenal syndrome (HRS) or renal failure defined as a serum creatinine  $> 221 \mu mol/L$  (> 2.5 mg/dL) or the requirement for renal replacement therapy;
- 14) Subjects dependent on inotropic (eg, epinephrine or norepinephrine) or ventilatory support (ie, endotracheal intubation or positive-pressure ventilation);
- 15) Portal vein thrombosis;
- 16) Acute pancreatitis;
- 17) Cessation of alcohol consumption for more than 2 months before Baseline/Day1;
- 18) Severe associated disease (eg, cardiac failure, acute myocardial infarction, severe cardiac arrhythmias, severe pulmonary disease, neurologic disease) that may lead to premature mortality within the study period;
- 19) Malignancy within the 2 years prior to Screening, with the exception of specific cancers that have been cured by surgical resection (eg, basal cell skin cancer). Subjects under evaluation for possible malignancy are not eligible;
- 20) Positive urine screen for amphetamines, cocaine or opiates (ie, heroin, morphine) at Screening. Subjects on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to Screening may be included in the study. Subjects with positive cannabis drug screen may be included in the study. Subjects with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator;
- 21) Treatment with immunosuppressive drugs [budesonide, tacrolimus, sirolimus, cyclosporine, azathioprine, mycophenolate mofetil, and methotrexate], pentoxifylline, N-acetylcysteine (NAC), or granulocyte (macrophage) colony-stimulating factor within 6 months of Screening. Subjects will be eligible to enroll if systemic corticosteroids were started within 3 days prior to the Baseline/Day 1 visit. Inhaled and topical corticosteroids are allowed;

- 22) Use of strong CYP3A4 inducers (eg carbamazepine, phenytoin, rifampin, St. John's wort) within 2 weeks of the Baseline/Day 1visit;
- 23) Active ocular herpes simplex;
- 24) Any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results;
- 25) Participation in another investigational study of a drug or device within 1 month prior or within 5 half-lives of the prior investigational agent (whichever is longer) prior to Screening;
- 26) Concurrent participation in another therapeutic clinical study;
- 27) Known hypersensitivity to the study drugs (GS-4997 and prednisolone), the metabolites, or formulation excipients;
- 28) Presence of any condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, such as history of substance abuse other than alcohol use or a psychiatric or medical condition;
- 29) Unavailable for follow-up assessment or concern for subject's compliance with the protocol procedures;

Study Procedures/ Frequency: Screening assessments should be completed within 14 days of Baseline/Day 1 visit. Eligibility will be based on local laboratory testing. Refer to Section 6.9.10 Screening Laboratory Assessments for additional details.

After the Screening period and a randomization visit at Baseline/Day 1, study visits will occur on Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24. At minimum, vital signs, physical examination (PE), HE and ascites assessment, safety laboratory tests, alcohol consumption, and concomitant medications will be done at every visit. AEs will be collected up to 30 days after the last dose of any study drug and SAEs will be collected throughout the study.

During the hospitalization period, subjects will be evaluated daily with assessments to include a review of adverse events, concomitant medications, study drug adherence, and a symptom-directed PE including assessments for ascites and HE. Findings based on these assessments and laboratory investigations obtained by treating physicians as part of routine care will be assessed by the investigator for triggers that may necessitate further evaluation and/or treatment discontinuation and managed per Section 7 of the protocol.

#### PPD

Screening assessments will include complete medical history, PE including vital signs, HE, ascites, hepatorenal syndrome (HRS) and infection assessment, laboratory assessments (hematology, chemistry, coagulation tests, HIV serology, hepatitis B and C serologies, and urinalysis), pregnancy tests (for females of child-bearing potential), liver biopsy, liver ultrasound, standard 12-lead ECG, chest x-ray, AUDIT / SADQ questionnaires, adverse events and concomitant medication assessment.

#### Recent gastrointestinal bleeding:

Gastrointestinal bleeding will be treated and the subject stabilized during the Screening period for at least 48 hours prior to randomization.

#### Sepsis:

All subjects will be screened for infection with chest radiography, urinalysis, urine culture, paracentesis with ascitic fluid (if clinically-detectable ascites is present) cell count, differential, and culture, and blood cultures (all laboratory and imaging tests performed locally). Sepsis will be defined as the presence of any positive culture or the requirement for initiation of antibiotics due to clinical or radiological signs of infection. Culture-negative pyrexia and leukocytosis on their own will not be regarded as signs of active sepsis since these findings are often seen in subjects with AH without infection. Subjects with evidence of sepsis should be treated according to the following guidelines:

• Spontaneous bacterial peritonitis (SBP): AASLD Practice Guidelines: Management of Adult Patients with Ascites Due to Cirrhosis: Update 2012. (http://www.aasld.org/publications/practice-guidelines-0#practice\_guidelines\_accordion-block-2). Minimum recommended duration of antibiotic treatment is 5 days, and repeat ascitic fluid analysis must show a greater than 50% reduction in the number of neutrophils prior to randomization. If the initial ascitic fluid culture was positive, a repeat ascitic fluid culture should be negative prior to randomization. Patients with SBP who also have a serum creatinine >1 mg/dL, blood urea nitrogen >30 mg/dL, or total bilirubin >4 mg/dL should also receive 1.5 g albumin per kg body weight within 6 hours of detection and 1.0 g/kg 2 days later.

- Urinary tract infection (UTI): American Urological
  Association Adult UTI Guidelines (2016)
  (https://www.auanet.org/education/adult-uti.cfm). Minimum
  recommended duration of antibiotic treatment is 5 days for
  uncomplicated UTI, 7 days for uncomplicated UTI in patients
  with diabetes, and 14 days for complicated UTI. If the initial
  urine culture is positive, patients must have a repeat urine
  culture that is negative prior to randomization.
- Other infections: Investigator's discretion.

Once the subject has been treated for infection for a minimum of 2 days, and the sepsis is deemed under control by the investigator, the subject may continue Screening and be randomized if eligible within the Screening period If the initial blood culture is positive, patients must have a repeat blood culture that is negative prior to randomization.

Eligible subjects will be randomized to one of the two treatment groups. Prior to initial dosing, required Baseline/Day 1 assessments will be performed and will include vital signs, PE, HE, ascites, HRS and infection assessment, laboratory assessments, pregnancy tests (for females of child-bearing potential), and review of adverse events, concomitant medication, CLDQ questionnaire and alcohol consumption.

PPD

While on study, subjects will undergo the following procedures and laboratory assessments:

- CLDQ questionnaire at Baseline/Day 1, Weeks 4 and 24
- Sparse PK Sampling at Baseline/Day 1 and at Weeks 1, 2 and 4
- Blood for Biomarkers at Screening, Baseline/Day 1, and at Weeks 1, 2, 4, 8, 12 and 24
- Urine collection for Biomarkers at Baseline/Day 1, and at Weeks 4 and 24
- ELF<sup>TM</sup> Test and LOXL2 at Baseline/Day 1 and at Weeks 4, 12 and 24
- FibroScan (if available and in subjects without ascites) at Baseline/Day 1 and at Weeks 4 and 24
- 12-lead ECGs at Screening, Baseline/Day 1, and at Weeks 4 and 8

- Blood glucose, insulin and lipid profile at Screening, Baseline/Day 1 and at Weeks 4, 12 and 24
- Hemoglobin A1c at Baseline/Day 1 and at Weeks 12, and 24
- Urine collection at Screening (for drug screen, pregnancy screen, and to rule out infection)
- Stool collection at Baseline/Day 1 and at Weeks 4 and 24.
- Intensive PK Sub-study

PPD

# Test Product, Dose, and Mode of Administration:

- Treatment Group A: GS-4997 18 mg (1 x 18 mg tablet) AND prednisolone 40 mg (4 x 10 mg tablets) both administered orally once daily; n=50-60 subjects
- Treatment Group B: GS-4997 placebo (1 tablet) AND prednisolone 40 mg (4 x 10 mg tablets) administered orally once daily; n=50-60 subjects

Up to 60 subjects per arm will be randomized in order to obtain 50 subjects in each arm for the full analysis set (ie, subjects randomized with histologically-proven severe AH who took at least one dose of study drug)

Treatment will be administered for 28 days inclusive of inpatient, and if applicable, outpatient periods.

# Reference Therapy:

Prednisolone 10 mg tablets will be used.

#### Criteria for Evaluation:

Safety:

Safety will be evaluated by examining the incidence of treatment emergent adverse events, including serious adverse events, clinical laboratory tests, ECGs, and vital signs.

An independent, external Data Monitoring Committee (DMC) that includes two hepatologists and a PhD statistician will convene prior to study start, once 20 subjects have been treated for 28 days, and every 3 months thereafter to monitor the study for safety events including SAEs, deaths, premature discontinuation of treatment for AEs, grade 3 and higher AEs, grade 3 and higher treatment-emergent laboratory abnormalities, and individual stopping criteria for GS-4997/placebo study drug (see Section 7.5). The DMC will also evaluate (based on an unblinded review of safety data) and monitor for trial stopping criteria (see Section 8.11).

Efficacy:

The biological activity of prednisolone and the combination of GS-4997 and prednisolone will be evaluated using clinical outcomes and biomarker variables.

Pharmacokinetics:

The plasma concentration of GS-4997 and its metabolite, GS-607509, will be determined. The plasma concentration of other GS-4997 metabolites and/or prednisolone may be explored. PK samples may also be used to measure protein-binding of GS-4997 and/or its metabolites. PPD

#### Statistical Methods:

#### **Primary Endpoint:**

The primary endpoint is the safety of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe AH. The primary analysis will be conducted when all subjects have been followed for 30 days after their last dose of study drug or been prematurely terminated from study.

#### Secondary Endpoints:

- Clinical outcomes
  - Mortality at 28 days, 8 weeks, 12 weeks, and 24 weeks
  - HRS
  - Infection
  - Length of hospital stay

- Liver transplantation
- Measures of hepatic synthetic function:
  - Change from baseline in liver biochemistry: ALT, AST, GGT, albumin, alkaline phosphatase, bilirubin, and INR
  - Lille response (score < 0.45) at Day 7, Lille null response (score ≥ 0.56) at Day 7, Lille score at Day 7 as a continuous variable, and combined score including Lille score at Day 7 and baseline MELD score
  - Change from baseline in prognostic indices: MELD, Child-Pugh score, Maddrey's DF

# **Exploratory Endpoints:**



#### **Efficacy Analysis:**



# **Exploratory Analysis:**

PPD

#### Safety Analysis:

All safety data collected will be listed and summarized, as appropriate, by treatment group. Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical variables or 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous variables by treatment group.

#### Pharmacokinetic Analysis:

GS-4997 and GS-607509 plasma concentrations will be listed and summarized for all subjects. PPD



#### Sample Size:

The number of subjects was chosen based on clinical experience with other similar proof-of-concept studies. PPD



This study will be conducted in accordance with the guidelines of Good Clinical Practice (GCP) including archiving of essential documents.

#### GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

° C degrees Celsius° F degrees FahrenheitADR adverse drug reaction

AE adverse event

AH Alcoholic Hepatitis

ALT alanine aminotransferase

ARA acid reducing agent

ASK1 apoptosis signal-regulating kinase 1

ASK1<sup>-/-</sup> apoptosis signal-regulating kinase 1 deficient

AST aspartate aminotransferase ATP Adenosine triphosphate

AUC<sub>tau</sub> area under the plasma concentration versus time curve over the dosing

interval (tau)

AUDIT Alcohol Use Disorders Identification Test β-hCG beta human chorionic gonadotropin

BAP Biomarker Analysis Plan

BMI body mass index
BUN blood urea nitrogen
CBC complete blood count
cc cubic centimeter
CI confidence interval
CK18 cytokeratin (C18)
CL<sub>cr</sub> creatinine clearance

C<sub>last</sub> last observed quantifiable plasma/serum concentration of the drug

C<sub>max</sub> maximum observed plasma/serum concentration of drug

CLDQ Chronic Liver Disease Questionnaire
CRO contract (or clinical) research organization

CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

CYP3A4 cytochrome P4503A
DKD Diabetic kidney disease

dL Deciliter

DMC Data Monitoring Committee

DSPH Drug Safety and Public Health

DF (Maddrey's) Discriminant Function

DP drug product
EC ethics committee
ECG electrocardiogram

Gilead Sciences, Inc. Amendment 3

eCRF electronic case report form **EDC** electronic data capture

example eg

ELF<sup>™</sup> Test enhanced liver fibrosis test

EoT **End of Treatment** EU European Union **FAS** Full analysis set

FDA (United States) Food and Drug Administration

FIO<sub>2</sub> Fraction of Inspired Oxygen **FSH** Follicle-stimulating hormone **GGT** gamma glutamyl transferase

GI gastrointestinal

**GMP** Good Manufacturing Practice

GSI Gilead Sciences, Inc. HbA1c Hemoglobin A1c

**HBsAg** Hepatitis B surface antigen

**HBV** Hepatitis B virus

**HCC** Hepatocellular Carcinoma hCG human chorionic gonadotropin

Hct Hematocrit **HCV** Hepatitis c virus

HDL High-density lipoprotein **HDPE** High-density polyethylene HE hepatic encephalopathy

Hg Hemoglobin

HIV Human immunodeficiency virus

HLT high-level term HLGT high-level group term

HOMA-IR homeostatic assessment of insulin resistance

HRS Hepatorenal Syndrome IΒ Investigator's Brochure **ICF** Informed Consent Form

International Conference on Harmonisation of Technical Requirements for **ICH** 

Registration of Pharmaceuticals for Human Use

ID Identification

**IEC** independent ethics committee **IEC** institutional ethics committee **IMP Investigational Medicinal Product** IND Investigational New Drug (Application)

**INR** international normalized ratio IRB institutional review board

IUDintrauterine deviceIVDIn vitro diagnostic

IWRS interactive web response system

kg Kilogram LOX Lysyl oxidase LOXL1 Lysyl oxidase-like 1 LOXL2 Lysyl oxidase-like 2 LOXL3 Lysyl oxidase-like 3 LOXL4 Lysyl oxidase-like 4 LPS lipopolysaccharide mAB monoclonal antibody

Medical Dictionary for Regulatory Activities

MELD Model for End-Stage Liver Disease

μg Microgram
mg Milligram
min Minute
mL Milliliter
mm Millimeter

mm Hg millimeters of mercury NAC N-acetylcysteine

NASH Nonalcoholic steatohepatitis
PAH Pulmonary arterial hypertension

PE Physical Exam
PK Pharmacokinetic

pH measure of the acidity

PT preferred term
PT prothrombin time
PTM Placebo to match

PTT Partial prothrombin time

q Every

QoL Quality of Life

QT electrocardiographic interval between the beginning of the Q wave and

termination of the T wave, representing the time for both ventricular

depolarization and repolarization to occur

RNA ribonucleic acid ROW rest of world

SADQ Severity of Alcohol Dependence Questionnaire

SADR serious adverse drug reaction

SAE serious adverse event

SAP statistical analysis plan

SBP Spontaneous bacterial peritonitis

SC Subcutaneous

SOP standard operating procedure

SUSAR Suspected Unexpected Serious Adverse Reaction

 $t_{\frac{1}{2}}$  An estimate of the terminal elimination half-life of the drug in

serum/plasma/PBMC, calculated by dividing the natural log of 2 by the

terminal elimination rate constant ( $\lambda_z$ )

TEAEs Treatment emergent adverse events

 $T_{last} \hspace{1cm} last \hspace{1cm} measured \hspace{1cm} concentration \\ T_{max} \hspace{1cm} time \hspace{1cm} (observed \hspace{1cm} time \hspace{1cm} point) \hspace{1cm} of \hspace{1cm} C_{max}$ 

TQT thorough QT

ULN upper limit of the normal range

US United States

UTI Urinary tract infection

wks weeks

#### 1. INTRODUCTION

# 1.1. Background

Alcoholic liver disease (ALD) encompasses a spectrum of disease ranging from reversible fatty liver to alcoholic hepatitis (AH) and cirrhosis. In the United States, ALD remains the second most common cause of liver cirrhosis after Hepatitis C virus (HCV) infection and is responsible for approximately 20% to 25% cases of liver cirrhosis {Gao 2011, Singal 2013}. In Western Europe, ALD is the most prevalent cause of advanced liver disease and cirrhosis is the leading cause of alcohol-related death among adults {European Association for the Study of the Liver (EASL) 2012}.

AH represents one of the most serious forms of ALD and remains a significant cause of morbidity and mortality in North America and Europe. Approximately 60% of patients with ALD in the United Kingdom will have evidence of an alcohol-related hepatitis at presentation {Hislop 1983}. In the United States (US), the burden of AH is increasing, with an estimated 326,000 hospitalizations (0.8% of all admissions) in 2010, a 30% increase compared with 2002 {Jinjuvadia 2015}. The mean length of a hospital stay is 5 to 7 days with an average health care cost of \$35,000 to \$41,000. In patients with severe AH (typically defined by a Maddrey's Discriminant Function (DF)  $\geq$  32, short-term mortality rates are high (approximately 25% to 45%) {Akriviadis 2000, Mathurin 2011}.

AH is a syndrome characterized by infiltration of the liver by inflammatory cells and hepatocellular injury. Several studies in rodent models and histopathological studies in humans suggest that lipopolysaccharide (LPS)-induced inflammation and oxidative stress are key drivers of hepatocyte death in AH {Chayanupatkul 2014, Lucey 2009, Meagher 1999}. Alcohol consumption increases intestinal permeability and bacterial translocation to the liver, resulting in LPS-induced hepatic inflammation. Subsequent hepatocellular injury occurs by neutrophil oxidative bursts, and FAS ligand and TNF- $\alpha$  induced hepatocyte apoptosis. In addition, ethanol strongly induces the expression of CYP2E1, which produces reactive oxygen species (ROS) as a by-product of ethanol metabolism, and reduces hepatic antioxidant capacity. Oxidative stress occurs as a result of these changes and directly induces hepatocyte mitochondrial dysfunction and necrosis and also sensitizes hepatocytes to apoptosis induced by TNF- $\alpha$  and FAS ligand {Cederbaum 2012}.

Pharmacologic agents that modulate these pathways have been used in the treatment of AH with limited success. Corticosteroid therapy which abrogates the inflammatory process is the current standard of care therapy for patients with severe AH. Compared with no treatment, a 28-day course of prednisolone improves 1-month mortality (approximately 35% vs. 20%), but shows limited impact on longer term outcomes {O'Shea 2010}. Indeed, 6-month mortality remains high despite prednisolone therapy {Mathurin 2011, Thursz 2015}. In addition to the limited efficacy of corticosteroids, there remains a high risk of infection in patients with severe AH who receive prednisolone {Louvet 2009}. In a cohort of 162 patients with AH (established by biopsy), 20% of patients had infections at hospital admission and 52% of those treated with corticosteroids

developed infections, including some patients with invasive aspergillosis {Michelena 2015}. In infected patients, the incidence of multiorgan failure (MOF, approximately 60%) and mortality (approximately 45% at 90 days) are substantially increased compared to uninfected patients (approximately 5% at 90 days). High-dose corticosteroids may also exacerbate glycemic control in diabetic patients and lead to an increased risk of gastrointestinal hemorrhage {Rudler 2015}. Other therapies that have been evaluated including pentoxifylline which modulates *TNF-α* transcription, N-acetylcysteine (an antioxidant), TNF inhibitors and antifibrotics, but none have shown convincing clinical benefit and/or are considered harmful {Mathurin 2011, Nguyen-Khac 2011, O'Shea 2005, Spahr 2002}. In light of the increasing burden of disease and limited therapeutic options, there remains a significant unmet medical need for alternative therapies with improved safety and efficacy for patients with severe AH.

#### 1.2. GS-4997

#### 1.2.1. General Information

GS-4997 is a small molecule that is a potent and selective inhibitor of apoptosis signal-regulating kinase 1 (ASK1). ASK1, a critical serine/threonine kinase, is an important signaling node through which oxidative stress promotes inflammation, proliferation, apoptosis, and fibrosis {Fujisawa 2007, Takeda 2008, Tobiume 2001, Watanabe 2005}. The ASK1 protein is ubiquitously expressed and is normally bound and repressed by thiol-containing antioxidant proteins in the cytosol and mitochondria {Fujino 2007, Takeda 2008, Zhang 2004}. In settings of elevated oxidative stress, ASK1 is autophosphorylated {Tobiume 2002}. The phosphorylated ASK1 then phosphorylates mitogen-activated protein kinase (MAPKKs) 3, 4, 6, and 7, which in turn phosphorylate and activate the mitogen-activated protein kinases (MAPKs) p38 and c-Jun N-terminal kinase (JNK) {Nagai 2007, Takeda 2008}.

In pathological settings of oxidative stress, ASK1 is required for sustained activation of p38 and JNK, which promotes the expression of inflammatory cytokines (eg, interleukins 1β, 2, and 6), chemokines (eg, monocyte chemotactic protein 1, chemokine ligands 1 and 2), and matrix remodeling genes (ie, transforming growth factor beta, tissue inhibitor of metalloproteinase, and plasminogen activator inhibitor-1) {Matsuzawa 2005, Mnich 2010, Nakamura 2009, Takeda 2008, Terada 2007, Tobiume 2001, Yokoi 2006}. Activation of the ASK1 pathway also increases the expression of nicotinamide adenine dinucleotide phosphate-oxidase and induces mitochondrial damage leading to an increase in the production of reactive oxygen species (ROS), apoptosis, necrosis, and in certain contexts, insulin resistance {Adachi 2013, Gerczuk 2012, Imoto 2006, Nakagawa 2008, Takeda 2008, Toldo 2012, Watanabe 2005}.

A potential role for ASK1 in AH is supported by nonclinical studies demonstrating that oxidative stress, Fas ligand and TNF-α signaling activate ASK1 in the mouse liver {Nakagawa 2011}. In addition,  $ASK1^{-/-}$  mice are resistant to acute liver injury caused by Fas activation, TNF-α (induced by LPS plus D-galactosamine), bile duct ligation, or acetaminophen overdose {Nakagawa 2011, Nakagawa 2008, Noguchi 2014}. Moreover, pharmacological inhibition of ASK1 in mice reduces hepatocellular injury and necrosis induced by acetaminophen overdose, as well as cardiac and renal apoptosis and necrosis induced by acute ischemia/reperfusion injury

{Toldo 2012, Xie 2015}. These effects correlated with reduced activation/phosphorylation of ASK1, p38, and JNK, and reduced mitochondrial dysfunction which could translate into improved liver function and resultant improved mortality in severe AH.

#### 1.2.2. Preclinical Pharmacology and Toxicology

GS-4997 has high oral bioavailability, moderate volume of distribution and low systemic clearance in nonclinical species and humans. GS-4997 is modestly bound in human plasma. Elimination of GS-4997 and its metabolites is likely to occur through a mixture of urinary, biliary and intestinal excretion. The main route of metabolism of GS-4997 involves N-dealkylation. Human metabolism appears to be largely catalyzed by cytochrome P4503A (CYP3A) enzymes. After oral dosing of GS-4997 significant concentrations of GS-607509, inactive N-dealkylation metabolite, are found in plasma. GS-4997 is an inhibitor of CYP3A and UDP glucuronosyltransferase family 1 member A1 (UGT1A1) enzymes; however, clinically relevant inhibition of CYP3A was not observed in humans. GS-4997 is a weak inhibitor of the transporters breast cancer resistance protein (BCRP), OATP1B1, and OATP1B3 and a more potent inhibitor of P-glycoprotein (P-gp), Organic cation transporter 1 (OCT1), Organic cation transporter 2 (OCT2), and Multidrug and toxin extrusion protein 1 (MATE1). The metabolite GS-607509 did not inhibit any of the CYP enzymes and was a very weak inhibitor of UGT1A1. GS-607509 shows little inhibition of all tested transporters apart from MATE1.

GS-4997 has been extensively evaluated in nonclinical toxicology studies. Findings attributed to GS-4997 administration were primarily related to the cardiovascular system (mild decrease blood pressure and mild QT interval corrected for heart rate (QTc) prolongation), GI tract (profuse diarrhea) and kidney (tubular basophilia, eosinophilic droplets, and pigment), embryofetal effects (visceral and/or skeletal malformations) and occurred at exposures that were in excess of the targeted human exposure at 18 mg/day. Similar findings have not been observed to date in clinical studies of GS-4997 at doses of up to 100 mg/day. Self-limiting diarrhea has been observed in subjects across the clinical studies. However, the low grade and self-limiting nature of the diarrhea suggests the diarrhea in the clinical studies is different from what was observed in monkeys.

Please refer to the GS-4997 IB for additional details.

#### 1.2.3. Clinical Trials of GS-4997

As of 14 October 2016, 13 Phase 1 and 2 clinical studies have been conducted/are ongoing in which 359 healthy subjects, 248 subjects with diabetic kidney disease (DKD), 113 subjects with pulmonary arterial hypertension (PAH), 72 subjects with NASH have been dosed with GS-4997.

Information on the completed and ongoing Phase 1 clinical studies can be found in the IB.

# 1.2.4. A Phase 2, Double-blind, Placebo-controlled, Dose-ranging Study Evaluating the Efficacy, Safety, and Tolerability of GS-4997 in Subjects with Diabetic Kidney Disease (Study GS-US-223-1015)

Study GS-US-223-1015 is an ongoing Phase 2, double-blind, placebo-controlled, dose-ranging study evaluating the efficacy, safety, and tolerability of GS-4997 in subjects with Diabetic Kidney Disease (DKD). Three-hundred and thirty-three subjects with type 2 diabetes mellitus and Stage 3 or Stage 4 renal impairment and albuminuria receiving standard of care treatment for DKD were randomized (1:1:1:1) to 1 of 4 treatment groups: GS-4997 2, 6, or 18 mg or matching placebo administered once daily for 48 weeks. The primary objective of this study is to determine the effect of GS-4997 on the decline of estimated glomerular filtration rate (eGFR) in subjects with DKD.

#### 1.2.4.1. Subject Disposition

Of the 334 randomized subjects, 333 subjects were treated with placebo or study drug: 85 subjects with placebo and 248 subjects with active treatment (81, 84, and 83 subjects with GS-4997 2, 6, and 18 mg, respectively).

A total of 256 subjects (76.9%) completed treatment and 76 subjects (22.8%) discontinued study drug (19 subjects [22.4%] in the placebo group and 57 subjects [23.0%] in the pooled active treatment group [18.5%, 21.4%, and 28.9% for GS-4997 2, 6, and 18 mg, respectively]). The most frequent reason for discontinuation of study drug was due to an AE (4 subjects [4.7%] in the placebo group and 18 subjects [7.3%] in the pooled active treatment group), followed by progression to end-stage renal disease (4 subjects [4.7%] in the placebo group and 13 subjects [5.2%] in the pooled active treatment group), and withdrawal of consent (3 subjects [3.5%] in the placebo group and 13 subjects [5.2%] in the pooled active treatment group).

#### 1.2.4.2. Preliminary Safety Analyses

Overall 80.8% of subjects had a treatment-emergent adverse event with a frequency of 83.5% in the placebo group and 79.8% in the pooled active group (79%, 84.5%, and 75.9% for 2 mg, 6 mg and 18 mg, respectively). Adverse events related to study drug occurred in 9.4% in placebo and 12.5% in the pooled active treatment group (8.6%, 11.9%, and 16.9% for 2 mg, 6 mg and 18 mg, respectively). Overall, deaths occurred in 1.2% of subjects with a frequency of 1.2% in the placebo group and 1.2% in the pooled active treatment group (1.2%, 1.2%, and 1.2% for 2 mg, 6 mg and 18 mg, respectively).

# 1.2.4.3. Preliminary Efficacy Analyses

The primary endpoint measure of eGFR change from baseline at Week 48 was -3.20 (SE 0.85), -2.83 (0.86), -2.37 (0.87), and -4.07 (0.89) mL/min/1.73 m<sub>2</sub> for placebo, 2 mg, 6 mg and 18 mg GS-4997 respectively (p= NS). The study did not demonstrate that GS-4997 led to a statistically significant decrease in eGFR after 48 weeks of treatment compared to placebo.

# 1.2.5. A Phase 2, Dose-ranging, Randomized, Double-blind, Placebo-controlled Study of GS-4997 in Subjects with Pulmonary Arterial Hypertension (Study GS-US-357-1394)

Study GS-US-357-1394 is an ongoing Phase 2, randomized, double-blind, placebo-controlled, multicenter, dose-ranging study of GS-4997 in subjects with PAH receiving background stable PAH therapy. One-hundred and fifty-one subjects with a diagnosis of idiopathic PAH (IPAH), heritable PAH (HPAH), or PAH associated with connective tissue disease (PAH-CTD), congenital heart defects (repaired), drug and toxin use, or HIV infection were randomized 1:1:1:1 to receive either GS-4997 2, 6, or 18 mg or placebo, orally, once daily, for 24 weeks. Subjects continued to receive their background PAH therapy throughout the study. Subjects who complete the 24-week blinded treatment period will be eligible to continue (or initiate) treatment with GS-4997 at 2, 6, or 18 mg during the blinded, long-term treatment extension of this study. The primary objective of this study is to evaluate the effect of GS-4997 on pulmonary vascular resistance (PVR), as measured by right heart catheterization (RHC) in subjects with PAH.

#### 1.2.5.1. Subject Disposition

Of the 151 randomized subjects, 150 subjects were treated with placebo or study drug: 37 subjects with placebo and 113 subjects with active treatment (39, 37, and 37 subjects with GS-4997 2, 6, and 18 mg, respectively).

A total of 134 subjects (89.3%) completed Period 1 treatment and 16 subjects (10.7%) discontinued study drug before reaching Week 24 (5 subjects [13.5%] in the placebo group and 11 subjects [9.7%] in the pooled active treatment group [10.3%, 13.5%, and 5.4% for GS-4997 2, 6, and 18 mg, respectively]). The most frequent reason for discontinuation of study drug was due to an AE (3 subjects [8.1%] in the placebo group and 6 subjects [5.3%] in the pooled active treatment group), followed by death (1 subject [2.7%] in the placebo group and 3 subjects [2.7%] in the pooled active treatment group), and investigator's discretion (2 subjects [1.8%] in the pooled active treatment group).

# 1.2.5.2. Preliminary Safety Analyses

Overall, 91.3% of subjects had a treatment-emergent adverse event with a frequency of 97.3% in the placebo group and 89.4% in the pooled active group (87.2%, 91.9%, and 89.2% for 2 mg, 6 mg and 18 mg, respectively). Adverse events related to study drug occurred in 48.6% in placebo and 42.5% in the pooled active treatment group (25.6%, 56.8%, and 45.9% for 2 mg, 6 mg and 18 mg, respectively). Overall, deaths occurred in 6.0% of subjects with a frequency of 8.1% in the placebo group and 5.3% in the pooled active treatment group (2.6%, 8.1%, and 5.4% for 2 mg, 6 mg and 18 mg, respectively).

# 1.2.5.3. Preliminary Efficacy Analyses

The primary efficacy endpoint was change in PVR from baseline to Week 24. The primary endpoint measure of median change in PVR from baseline to Week 24 was -43 (CI -99, 86), 23 (-45, 146), -39 (-97, 36) and -40 (-74, -7) dynes\*sec/cms for placebo, 2 mg, 6 mg and 18 mg GS-4997, respectively (p=0.36). The study thus did not demonstrate that GS-4997 led to a statistically significant change in PVR after 24 weeks of treatment compared to placebo.

1.2.6. A Phase 2, Randomized, Open Label Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 alone or in Combination with Simtuzumab (SIM) in Subjects with Nonalcoholic Steatohepatitis (NASH) and Fibrosis (F2-F3) (GS-US-384-1497)

This multicenter, randomized, open-label study evaluated the safety, tolerability, and efficacy of GS-4997 (6 mg or 18 mg) alone or in combination with simtuzumab (SIM, a monoclonal antibody directed against LOXL2 evaluated for the treatment of NASH) for 24 weeks in subjects with NASH and fibrosis stages F2 or F3.

The primary objective of this study was to evaluate the safety and tolerability of GS-4997 alone or in combination with SIM in subjects with NASH and fibrosis stages F2 or F3.

Subjects were randomized in a 2:2:1:1:1 ratio to 1 of 5 treatment groups:

- GS-4997 6 mg orally once daily (N = 20)
- GS-4997 18 mg orally once daily (N = 22)
- GS-4997 6 mg orally once daily + SIM 125 mg subcutaneous injection weekly (N = 10)
- GS-4997 18 mg orally once daily + SIM 125 mg subcutaneous injection weekly (N = 10)
- SIM 125 mg subcutaneous injection weekly (N = 10)

Overall, after 24 weeks of treatment, no additional benefit was observed with the addition of SIM 125 mg to the GS-4997 (18 or 6 mg) study treatment regimens. Moreover, data from the SIM Phase 2b program (studies GS-US-321-0105 and GS-US-321-0106) showed that SIM has no anti-fibrotic effect in subjects with advanced fibrosis due to NASH. Therefore, preliminary efficacy results are presented by the following pooled groups: GS-4997 18 mg  $\pm$  SIM 125 mg, GS-4997 6 mg  $\pm$  SIM 125 mg, and SIM 125 mg alone.

#### 1.2.6.1. Subject Disposition and Demographics

A total of 72 subjects were randomized and treated across 23 sites (21 in the US and 2 in Canada); 67 subjects (93.1%) completed study treatment. Of the 5 subjects who did not complete study treatment, 3 subjects discontinued due to AEs, 1 subject withdrew consent, and 1 subject was lost to follow-up.

# 1.2.6.2. Preliminary Safety Results

Overall, 79.2% of subjects had a treatment-emergent adverse event with a frequency of 70% in the SIM alone group and 80.6% in the pooled active group (85%, 68.2%, 90%, and 90% in the GS-4997 6 mg, GS-4997 18 mg, GS-4997 6 mg + SIM, and GS-4997 18 mg + SIM, respectively). Adverse events related to study drug occurred in 0% of the SIM alone group and 33.9% in the pooled active treatment group (40%, 31.8%, 20%, and 40% in the GS-4997 6 mg, GS-4997 18 mg, GS-4997 6 mg + SIM, and GS-4997 18 mg + SIM, respectively).

Overall, GS-4997 6 mg or 18 mg ± SIM 125 mg administered for 24 weeks was generally well tolerated in study GS-US-384-1497. The majority of subjects reported at least 1 AE, and most AEs were mild or moderate in severity. Three subjects discontinued study treatment due to AEs: 2 subjects (9.1%) in the GS-4997 18 mg group (diarrhea and hypoesthesia in 1 subject and increased hepatic enzymes in 1 subject) and 1 subject (5.0%) in the GS-4997 6 mg group (worsened schizophrenia). A total of 11 SAEs were reported in 5 subjects during the study. Of these, only 1 SAE (hypoesthesia) was considered related to study drug by the investigator. No trends in SAE type or onset were observed. There were no deaths reported. Treatment-emergent Grade 3 and 4 laboratory abnormalities were infrequent. There were 4 subjects who developed an increase of ALT or AST of at least 2 × Baseline and at least 3 × ULN, leading to permanent discontinuation of study drug in 1 subject. No trends in ECG findings suggestive of cardiac abnormalities were observed.

# 1.2.6.3. Preliminary Efficacy Results

Subjects treated with GS-4997 (18 or 6 mg)  $\pm$  SIM 125 mg had a  $\geq$  1-stage decrease in NASH CRN fibrosis stage from baseline in 43.3% and 29.6% of subjects, respectively, compared with 20.0% of subjects treated with SIM 125 mg alone. Subjects treated with GS-4997 (18 or 6 mg)  $\pm$  SIM 125 mg were less likely to have worsening of fibrosis (6.7% and 14.8%, respectively) or progression to cirrhosis (3.3% and 7.4%, respectively) compared with subjects treated with SIM 125 mg alone (40.0% with worsening of fibrosis and 20.0% with progression to cirrhosis).

For further information on GS-4997, refer to the IB for GS-4997.

#### 1.3. Rationale for This Study

ASK1 is a serine/threonine kinase that is activated by oxidative stress and stimulates apoptotic, fibrogenic, and inflammatory pathways via p38 and JNK activation. In mouse models of non-alcoholic acute liver injury, ASK-1 has been shown to promote hepatocyte apoptosis and necrosis {Nakagawa 2011}. In an internal study, liver biopsies from 9 patients with severe AH were shown to have significantly higher p-p38 immunoreactivity (an indicator of ASK1 pathway activation) compared to biopsies from patients with NASH and PSC suggesting that ASK1 inhibition may be a potential therapeutic target in severe AH. GS-4997 is a small molecule, potent and selective inhibitor of ASK1. Inhibition of ASK1 with GS-4997 and resultant reduction of oxidative stress-induced hepatocyte apoptosis and necrosis, which are key mediators of AH pathogenesis {Ziol 2001} is hypothesized to improve efficacy and safety

compared with corticosteroid treatment in patients with AH. Moreover, data from the Phase 2 study GS-US-384-1497 in patients with NASH and moderate to severe fibrosis that demonstrated an anti-fibrotic effect of GS-4997 (18 mg or 6 mg daily  $\pm$  SIM) support its evaluation in patients with severe AH, the majority of whom have advanced fibrosis.

Mortality in AH is associated with acute loss of liver function and accompanying complications of advanced liver disease, including encephalopathy, sepsis, and/or MOF including renal failure. Data generated at Gilead have demonstrated that ASK1 inhibition does not directly reduce LPS-mediated signaling and cytokine release by macrophages, nor does it reduce oxidative burst by neutrophils. These pathways are considered important mechanisms in the pathophysiology of severe AH. However it is hypothesized that the hepatoprotective effects of GS-4997 via other mechanisms could translate into improved liver function and resultant improved mortality in severe AH. Early improvement in liver function is associated with better survival (eg. 1-6 months following presentation) {Louvet 2015, Louvet 2007}. Prednisolone is the standard of care for severe AH and has been shown to reduce systemic levels of cytokines (ie, TNF- $\alpha$ , IL-8) and reduce neutrophil activity (oxidative burst) in patients with severe AH {Taieb 2000}. The complementary mechanisms of action of GS-4997 and prednisolone suggest a potential benefit could be gained via their combination. Given the distinct mechanism of action of GS-4997 and the totality of the preclinical evidence of modulating pathways involved in liver damage in AH, evaluating the combination of GS-4997 and prednisolone in patients with AH is of merit.

#### 1.4. Rationale for Dose Selection

GS-4997 tablets will be administered orally once daily at a dose of 18 mg.

In preclinical models of DKD, PAH, NASH, and acute acetaminophen overdose, maximal efficacy is achieved with a dose that provides near complete suppression of the ASK1 pathway in target tissues (> EC95). For this Phase 2 proof-of-concept study, the dose selected (18 mg once daily) is projected to provide a plasma concentration that is expected to cause near complete inhibition of ASK1 (> EC95) at trough based on an ex vivo CXCL1 assay in human whole blood (CXCL1 EC95 = 130 ng/mL) to maximize potential for efficacy in this severe acute indication. This dose selection is supported by a preliminary review of unblinded biomarker data from an ongoing double-blind Phase 2 study in DKD (GS-US-223-1015) evaluating doses of 2 mg, 6 mg, and 18 mg of GS-4997 once daily. Moreover, data from the Phase 2 study GS-US-384-1497 in patients with NASH and moderate to severe fibrosis demonstrated a numerically greater likelihood of fibrosis regression in subjects treated with 18 mg versus 6 mg of GS-4997 daily.

GS-4997 has been evaluated at doses up to 100 mg in Phase 1 studies and up to 18 mg in Phase 2 studies and, based on currently available blinded and unblinded safety data, is well tolerated. Based on in vitro and in vivo DDI results with probe drugs, GS-4997 PK is not expected to be significantly altered when coadministered with prednisolone as planned for this Phase 2 study. In the Phase 1 hepatic impairment study (GS-US-223-1018), there were minimal to modest changes in GS-4997 PK across varying degrees of hepatic impairment (mild, moderate, and severe). A 43% increase in GS-4997 exposure (AUC) in subjects with severe hepatic impairment is less than what was observed in Study GS-US-223-1434 with the strong CYP3A4 inhibitor ritonavir

(79% increase). The small increase in exposure observed with severe hepatic impairment is not considered clinically meaningful as the observed changes are less than or comparable to the expected effect of a moderate CYP3A4 inhibitor on GS-4997 exposure; moderate and strong CYP3A4 inhibitors are currently allowed in ongoing Phase 2 and Phase 3 studies evaluating doses of GS-4997 of up to 18 mg once daily. Based on the current safety/tolerability profile for GS-4997 at doses more than 5-fold higher than the dose proposed for this study, the increase in GS-4997 exposure in subjects with severe hepatic impairment is not considered clinically relevant and does not require dose adjustment. Taken together, these data support evaluation of GS-4997 18 mg once daily in subjects with severe AH.

# 1.5. Risk/Benefit Assessment for the Study

The primary risk of study participation relates to the proposed initiation of prednisolone  $\pm$  GS-4997 prior to the histologic confirmation of AH. The rationale for this approach is two-fold. First, in many centers, performance of liver biopsy in subjects with suspected severe AH is not standard of care prior to initiating treatment, typically with prednisolone. Second, the planned approach will allow the rapid initiation of therapy which is deemed vital to optimize outcomes in subjects with severe AH. Importantly, a clinical diagnosis of AH (as per standard of care) will be made and contraindications to prednisolone (e.g. untreated infection) will be excluded in all subjects prior to starting treatment.

Another related risk of study participation is that some subjects who do not have alcoholic hepatitis will be exposed to prednisolone  $\pm$  GS-4997 therapy for up to 7 days before the diagnosis is refuted on biopsy. Based on prior studies, an estimated 20% of subjects who are suspected of severe alcoholic hepatitis do not have confirmation of the diagnosis on biopsy. As mentioned above, the initiation of prednisolone in subjects with suspected alcoholic hepatitis without performance of a liver biopsy is standard practice in many centers. The plan to discontinue treatment in subjects in whom the biopsy does not confirm alcoholic hepatitis is a potential benefit of study participation because it will limit exposure to prednisolone, which has toxicities including infection and worsened glycemic control The risk of short-term exposure to GS-4997 is low based on the results of prior Phase 1 and 2 studies (as outlined in Section 1.2.3), including the hepatic impairment study (GS-US-223-1018) that included subjects with mild, moderate, and severe hepatic dysfunction.

In view of the potential for GS-4997 to reduce major mechanisms of liver injury in subjects with severe alcoholic hepatitis, the limitations in available therapy, existing safety data, and the proposed study design to carefully monitor patient safety, the benefit/risk balance for this study is considered positive.

#### 1.6. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

# 2. OBJECTIVES

The primary objective of this study is:

 To evaluate the safety and tolerability of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe AH

The secondary objectives of this study are as follows:

- To assess changes in hepatic synthetic function [liver biochemistry, Model for End-Stage Liver Disease [MELD] score, Child-Pugh score, the Lille model, and Maddrey's Discriminant Function (DF)];
- To assess mortality at 28 days, Week 8, Week 12 and Week 24
- To determine the incidence of liver transplantation;
- To determine the incidence of hepatorenal syndrome (HRS);
- To determine the incidence of infection;
- To assess length of hospital stay;

The exploratory objectives of this study are:





# 3. STUDY DESIGN

# 3.1. Study Design

The overall study design is presented graphically in Figure 3-1.



<sup>\*</sup> Up to 60 subjects will be randomized leading to 50 subjects in each arm for the full analysis set (ie, histologically-proven severe AH and took at least one dose of study drug)

# 3.2. Treatment Plan and Regimen

This is a Phase 2 double blind, randomized study evaluating the safety, tolerability, and biological activity of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe, histologically-confirmed AH.

Up to 120 subjects will be randomized in a 1:1 ratio (within strata) to 1 of 2 treatment groups:

- Group A (n = 50-60): GS-4997 18 mg once daily + prednisolone 40 mg once daily for 28 days
- Group B (n = 50-60): GS-4997 placebo once daily + prednisolone 40 mg once daily once daily for 28 days

Randomization will be stratified by MELD < 25 or  $\ge 25$  at Screening as calculated using local laboratory tests and an online MELD calculator (see Section 6.9.7).

The full analysis set will comprise 100 subjects but up to 120 subjects will be randomized to account for subjects in whom AH is not confirmed on liver biopsy. The full analysis set includes those randomized and dosed with histologically-proven severe AH. Safety data will be reported for all subjects who take study drug.

All subjects with liver biopsies consistent with severe AH and negative HBV, HCV, and HIV serologies who complete study drug should complete Screening, on-treatment, and post-treatment assessments as outlined in Appendix 2. Subjects discontinuing both study drugs prior to Week 2 should complete an end of treatment visit after stopping drug, a 30-day safety FU visit, and all post-treatment follow-up visits. Subjects discontinued after Week 2 should complete an end of treatment visit, and all post-treatment assessments as outlined in Appendix 2.

Subjects whose liver biopsy results are not consistent with AH or whose HIV or hepatitis B or C serologies from the central laboratory are positive must stop study drug within 3 days of receipt of results. In subjects in whom a liver biopsy is insufficient to confirm a diagnosis of AH, subjects may remain in the study if no alternative diagnosis is suggested on biopsy. Subjects whose serum pregnancy testing from the central laboratory is positive at Screening must stop study drug immediately upon receipt of this result. All subjects stopping study drug for inconsistent liver biopsy results, for positive HIV or hepatitis B or C serologies from the central laboratory, or for positive serum pregnancy testing from the central laboratory should attend an EoT visit as soon as possible and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study (see Sections 6.7 and 6.8 of this protocol for clarification on study drug vs. study discontinuation).

#### **Intensive PK Sub-study**

PPD

#### 3.3. Biomarker Testing

# 3.3.1. Biomarker Samples to Address the Study Objectives

PPD

Stool samples may be used for microbiome analysis. The specific analyses will include, but will not be limited to, the biomarkers and assays listed below in Table 3-1. Because biomarker science is a rapidly evolving area of investigation, and adverse events in particular are difficult to predict, it is not possible to specify prospectively all tests that will be done on the specimens provided. The testing outlined is based upon the current state of scientific knowledge. It may be modified during or after the end of the study to remove tests no

longer indicated and/or to add new tests based upon the growing state of the art knowledge. If a test will no longer be performed because the assay is not robust, sample collection may also be withdrawn to reduce burden on subjects.

Specimens will be collected from all subjects. Samples will be destroyed no later than 15 years after the end of the study. The specimen storage period will be in accordance with the IRB/IEC/EC-approved Informed Consent Form (ICF) and applicable laws (eg, health requirements).

Table 3-1. Biomarkers

| Biomarker Focus | Planned Biomarkers | Rational | Specimen Collected |
|---|---|---|---|
| Liver tissue surrogate marker panel | ELF Test | Assess potential changes in liver fibrosis due to treatment | Blood |
| Liver tissue damage<br>marker | Serum LOXL2 | Assess potential changes in liver tissue damage due to treatment | Blood |
| Apoptosis and Necrosis markers | Circulating Cytokeratin 18<br>(CK18) fragments, M30<br>for apoptosis and M65 for<br>all dying cells) | Determine changes in liver cell death due to treatment | Blood |
| Inflammatory involvement | Serum cytokines | Determine changes in the inflammatory status due to treatment | Blood |
| Infection | Lipopolysaccharide<br>(LPS)/endotoxin | Assess changes in gut<br>barrier function due to<br>treatment | Blood |
| Infection | Procalcitonin | Assess changes in gut barrier function due to treatment | Blood |
| Metabolome | Circulating metabolite profiles (open platform) | Assess changes in the metabolome due to treatment | Blood |
| ASK1 pathway activity | phospho-p38* | blood marker of ASK1<br>pathway activity to<br>monitor PD effects | Blood |
| Intestinal microbial composition | Stool microbiome<br>determined by 16S<br>ribosomal DNA<br>sequencing | Assess changes in microbial populations due to treatment | Stool |
| ASK1 pathway activity | Focused panel gene expression (Nanostring) | Assess gene expression in disease at baseline | Liver Biopsy |
| ASK1 pathway activity | phospho-p38 IHC | Assess ASK1 pathway activation at baseline | Liver Biopsy |
| Biomarker Focus | Planned Biomarkers | Rational | Specimen Collected |
|---|---|---|---|
| FXR Pathway Activity | FGF19 | Assess FXR pathway activity to inform potential combinations | Blood |
| Urine biomarkers | Metabolite profile | Assess changes in biomarkers due to treatment not detected in blood | Urine |
| Circulating bacterial DNA | Bacterial DNA | Assess circulating bacterial DNA composition | Blood |
| Circulating Micro RNA | Serum miRNA | Assess changes in circulating miRNA associated with liver disease due to treatment | Blood |

<sup>\*</sup> Biomarker blood sample phospho-p38 will occur at US study sites.

For sampling procedures, storage conditions, and shipment instructions, see the Central Laboratory Services Manual.

# 3.3.2. Biomarker Samples for Optional Future Research





PPD

## 4. SUBJECT POPULATION

# 4.1. Number of Subjects and Subject Selection

The full analysis set will comprise 100 subjects, males and non-pregnant, non-lactating females between 18-70 years of age with histologically-confirmed severe AH (Maddrey's DF  $\geq$  32). Up to 20 additional subjects will be randomized to account for subjects in whom AH is not histologically-confirmed.

#### 4.2. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

- 1) Males and non-pregnant, non-lactating females between 18-70 years of age, inclusive based on the date of the Screening visit;
- 2) Willing and able to give informed consent prior to any study specific procedures being performed. In subjects with HE, which may impair decision-making, consent will be obtained per hospital procedures (eg, by legal Authorized Representative);
- 3) Clinical diagnosis of severe AH based on all of the following:
  - a) History of excessive alcohol consumption during the past 3 months (average of > 40 g/d of alcohol for women and > 50 g/d for men);
  - b) Aspartate aminotransferase (AST)  $\geq$  50 U/L, based on local laboratory results;
  - c) AST/alanine aminotransferase (ALT) ratio (AST/ALT) ≥ 1.5, based on local laboratory results;
  - d) Onset of jaundice within the past 3 months;
  - e) Maddrey's DF  $\geq$  32 at Screening, based on local laboratory results;
- 4) All female subjects of childbearing potential must agree to use a highly effective method of contraception during intercourse from the Screening visit throughout the study period and for 90 days following the last dose of study drug. If females utilize hormonal agents as one of their contraceptive methods, the same hormonal methods must have been used for at least 3 months before study dosing. Females on hormonal methods must also utilize a barrier method as another form of contraception as described in Appendix 3;
- 5) Male subjects must refrain from sperm donation from Screening through at least 90 days following the last dose of study drug;

- 6) Male subjects must agree to use condoms during intercourse from Screening through study completion and for 90 days following the last dose of study drug;
- 7) Female subjects must refrain from egg donation or harvest for 90 days after last dose of study drug;
- 8) Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions

#### 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study.

- 1) Pregnant or lactating females;
- 2) Other causes of liver disease including chronic hepatitis B (hepatitis B surface antigen [HBsAg] positive), chronic hepatitis C (HCV RNA positive), acetaminophen hepatotoxicity, biliary obstruction, and autoimmune liver disease
- 3) Serum AST > 400 U/L or ALT > 300 U/L, based on local laboratory results;
- 4) MELD > 30 at Screening, based on local laboratory results;
- 5) Maddrey's DF > 60 at Screening, based on local laboratory results;
- 6) Grade 4 HE by West Haven criteria;
- 7) Concomitant or previous history of hepatocellular carcinoma;
- 8) History of liver transplantation;
- 9) HIV Ab positive;
- 10) Clinical suspicion of pneumonia;
- 11) Uncontrolled sepsis;
- 12) Uncontrolled gastrointestinal (GI) bleeding or controlled GI bleeding within 7 days of Screening that was associated with shock or required transfusion of more than 3 units of blood;
- 13) Type 1 hepatorenal syndrome (HRS) or renal failure defined as a serum creatinine  $>221 \mu mol/L$  (> 2.5 mg/dL) or the requirement for renal replacement therapy;
- 14) Subjects dependent on inotropic (eg, epinephrine or norepinephrine) or ventilatory support (ie, endotracheal intubation or positive-pressure ventilation);

- 15) Portal vein thrombosis;
- 16) Acute pancreatitis;
- 17) Cessation of alcohol consumption for more than 2 months before Baseline/Day 1;
- 18) Severe associated disease (eg, cardiac failure, acute myocardial infarction, severe cardiac arrhythmias, severe pulmonary disease, neurologic disease,) that may lead to premature mortality within the study period;
- 19) Malignancy within the 2 years prior to Screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible.
- 20) Positive urine screen for amphetamines, cocaine or opiates (ie, heroin, morphine) at Screening. Subjects on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to Screening may be included in the study. Subjects with positive cannabis drug screen may be included in the study. Subjects with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator;
- 21) Treatment with immunosuppressive drugs [budesonide, tacrolimus, sirolimus, cyclosporine, azathioprine, mycophenolate mofetil, and methotrexate], pentoxifylline, N-acetylcysteine (NAC), or granulocyte (macrophage) colony-stimulating factor within 6 months of Screening. Subjects will be eligible to enroll if systemic corticosteroids were started within 3 days prior to the Baseline/Day 1 visit. Inhaled and topical corticosteroids are allowed;
- 22) Use of strong CYP3A4 inducers (eg, carbamazepine, phenytoin, rifampin, St. John's Wort) within 2 weeks of the Baseline/Day 1 visit;
- 23) Active ocular herpes simplex;
- 24) Any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the subject or impair the assessment of study results;
- 25) Participation in another investigational study of a drug or device within 1 month prior or within 5 half-lives of the prior investigational agent (whichever is longer) prior to Screening;
- 26) Concurrent participation in another therapeutic clinical study;
- 27) Known hypersensitivity to the study drugs (GS-4997 and prednisolone), the metabolites, or formulation excipient;

- 28) Presence of any condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, such as history of substance abuse other than alcohol use or a psychiatric or medical condition;
- 29) Unavailable for follow-up assessment or concern for subject's compliance with the protocol procedures.

# 5. INVESTIGATIONAL AND NON-INVESTIGATIONAL MEDICINAL PRODUCTS

## 5.1. Randomization, Blinding and Treatment Codes

This is a randomized, double blind study. An Interactive Web Response System (IWRS) will be used for centralized randomization and treatment assignment. Randomization will be stratified by MELD < or ≥ 25 at Screening as calculated using local laboratory tests and an online MELD calculator (see Section 6.9.7). Within each of the strata, subjects will be randomized in a 1:1 ratio to receive GS-4997 + prednisolone or GS-4997 placebo + prednisolone. Investigative site personnel will obtain the subject's identification number and study drug assignment from the IWRS. Study drug will be dispensed by the study pharmacist, or designee.

## 5.1.1. Procedures for Breaking Treatment Codes

In the event of a medical emergency where breaking the blind is required to provide medical care to the subject, the investigator may obtain treatment assignment directly from the IWRS system for that subject. Gilead recommends but does not require that the investigator contacts the Gilead medical monitor before breaking the blind. Treatment assignment should remain blinded unless that knowledge is necessary to determine subject emergency medical care. The rationale for unblinding must be clearly explained in source documentation and on the electronic case report form (eCRF), along with the date on which the treatment assignment was obtained. The investigator is requested to contact the Gilead medical monitor promptly in case of any treatment unblinding.

Blinding of study treatment is critical to the integrity of this clinical trial and therefore, if a subject's treatment assignment is disclosed to the investigator, the subject will have study treatment discontinued. All subjects will be followed until study completion unless consent to do so is specifically withdrawn by the subject.

Gilead Drug Safety and Public Health (DSPH) may independently unblind cases for expedited reporting of suspected unexpected serious adverse reactions (SUSARs).

## 5.2. Description and Handling of Study Drugs

#### 5.2.1. Formulation

# 5.2.1.1. GS-4997 18 mg and GS-4997 Placebo to Match (PTM)

GS-4997 will be supplied as 18 mg strength round, plain-faced, white film-coated tablets. In addition to the active ingredient, GS-4997 tablets contain the following commonly used inactive ingredients:

The matching placebo tablets are identical in physical appearance and contain the same inactive ingredients as the GS-4997 18 mg tablets.

## 5.2.1.2. Prednisolone

Commercially available prednisolone will be used for the study. Further information regarding formulation is available in the Prescribing Information for commercial product.

## 5.2.2. Packaging and Labeling

# 5.2.2.1. GS-4997 18 mg and GS-4997 PTM

GS-4997 18 mg and GS-4997 PTM tablets are packaged in white high density polyethylene (HDPE) bottles. Each bottle contains 30 tablets, silica gel desiccant and polyester packing material. Each bottle is enclosed with a white, continuous-thread, child-resistant polypropylene screw cap with an induction-sealed and aluminum-faced liner.

Study drug to be distributed to centers in the US and other participating countries shall be labeled to meet applicable requirements of the United States Food and Drug Administration (FDA), EU Guideline to Good Manufacturing Practice - Annex 13 (Investigational Medicinal Products), and/or other local regulations.

## 5.2.2.2. Prednisolone

Commercially available prednisolone 10 mg tablets will be used for the study.

## 5.2.3. Storage and Handling

### 5.2.3.1. GS-4997 and GS-4997 PTM

GS-4997 18 mg and GS-4997 PTM tablets should be stored at controlled room temperature of 25°C (77 °F); excursions are permitted between 15 °C and 30 °C (59 °F and 86 °F). Storage conditions are specified on the label. Until dispensed to the subjects, all bottles of study drug should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability and proper identification, study drug should not be stored in containers other than the containers in which they were supplied.

Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure when handling.

#### 5.2.3.2. Prednisolone

Commercially available prednisolone 10 mg tablets will be used for the study. Further information regarding storage and handling are available in the Prescribing Information for commercial product.

# 5.3. Dosage and Administration of Study Drugs

### **5.3.1. GS-4997**

GS-4997 18 mg and GS-4997 PTM tablets will be provided by Gilead Sciences. Once daily, at approximately the same time each morning, the study drug should be taken orally with water, swallowed whole, and with or without food. A dose will be considered missed if the subject cannot take the dose within 8 hours of their regular dosing time. If a subject misses a dose, the subject should take their next dose at the regular dosing time. For subjects who initiate dialysis, GS-4997/PTM should be administered following dialysis on days of the procedure and at the usual time on non-dialysis days. Please note that study drug should not be taken on mornings of sparse PK and biomarker assessments as outlined in Appendix 2. The dose should be taken as soon as possible after the trough PK and trough biomarker assessments are completed.

#### 5.3.2. Prednisolone

Commercially available prednisolone 10 mg tablets will be provided by Gilead Sciences. Subjects will take 40 mg prednisolone (4 x 10 mg) orally with water, once a day, with or without meals. The study drug should be swallowed whole and taken at approximately the same time each day. A dose will be considered missed if the subject cannot take the dose within 8 hours of their regular dosing time. The timing of prednisolone dosing should remain unchanged in subjects on dialysis. If a subject misses a dose, the subject should take their next dose at the regular dosing time. Prednisolone administration will not exceed 28 days from Baseline/Day 1 (a tapering course of prednisolone after the 28-day treatment period will not be allowed).

## 5.4. Prior and Concomitant Medications

*In vitro* data suggests that GS-4997 has the potential to inhibit P-glycoprotein (P-gp). GS-4997 has the potential to increase the exposure of sensitive P-gp substrates (eg, aliskiren, dabigatran etexilate, digoxin, fexofenadine, ranolazine). In a drug-drug interaction study of GS-4997 co-administered with digoxin (0.5 mg), exposure of digoxin (AUC) was increased by less than 30%. GS-4997 may increase the exposure of other P-gp substrates; however, the clinical relevance of such interactions has not been determined. Co-administration of P-gp substrates with study drug is allowed, with specific guidance provided for the following:

- Digoxin: Follow digoxin level at baseline and at the Week 1 visit with digoxin level checks during the study period per investigator discretion (as frequently as needed).
- Dabigatran etexilate: Consult Medical Monitor
- Ranolazine: Monitor for side effects
- Aliskiren: Use with caution, dose may need to be reduced

All concomitant medication will be recorded in the source documents. This includes concomitant medications taken within 30 days prior to Screening and any taken during the study to the end of

the follow-up period. Enteral and parenteral nutritional products administered during the study will be recorded on eCRFs.

### 5.5. Prohibited Medications

The use of any investigational medication or device in the 30 days prior to Screening and through the study is prohibited. Administration of pentoxifylline, NAC, or granulocyte (macrophage) colony-stimulating factor is prohibited within 6 months of Screening and through the study. Systemic corticosteroids are allowed only if administered within 3 days of Baseline/Day 1.



Co-administration of strong CYP3A4 inducers may decrease GS-4997 exposures. In a drug-drug interaction study of GS-4997 co-administered with repeat dose rifampin (strong CYP3A4 inducer), GS-4997 exposures were significantly reduced. Therefore, co-administration of strong CYP3A4 inducers (e.g. carbamazepine, phenytoin, rifampin, St. John's wort) with study drug is prohibited.

Examples of representative medications that are prohibited or which should be used with caution from 30 days prior to Day 1 through the treatment period are listed below in Table 5-1

Table 5-1. List of Prohibited Medications

| Drug Class | Agents Disallowed phenobarbital, phenytoin, carbamezepine, oxcarbazepine |
|---|---|
| Anticonvulsants <sup>a</sup> | |
| Antimycobacterials <sup>a</sup> | rifampin, rifabutin, rifapentine |
| Herbal/Natural<br>Supplements | St. John's Wort <sup>a</sup> , Echinaccea <sup>a</sup> , milk thistle (i.e. silymarin) <sup>a</sup> , Chinese herb sho-saiko-to (or Xiao-Shai-Hu-Tang) <sup>a</sup> |
| Immunosuppressants <sup>b</sup> | budesonide, tacrolimus, sirolimus, cyclosporine, azathioprine, mycophenolate mofeti<br>and methotrexate |
| Other <sup>c</sup> | Corticosteroids, pentoxifylline, N-acetylcysteine (NAC), or granulocyte (macrophage colony-stimulating factor |
| Drug Class | Agents to be used with Caution |
| Cardiac Medications | Digoxin <sup>e</sup> , ranolazine, dabigatran etexilate, aliskiren |

- a May result in a decrease in the concentration of GS-4997.
- b Prohibited within 6 months of Screening and through study.
- c Prohibited within 6 months of Screening and through study. Subjects will be eligible to enroll if systemic corticosteroids were started within 3 days prior to the Baseline/Day 1 visit. Inhaled and topical corticosteroids are allowed.
- d GS-4997 may increase the exposure of these medications.
- e For subjects on digoxin at start of study: obtain digoxin level prior to starting study drug and at the Week 1 Visit with digoxin level checks during the study period per investigator discretion. Monitor and adjust digoxin dose as necessary based on prescribing information.

# 5.6. Study Drug Accountability

The investigator or designee (eg, pharmacist) is responsible for ensuring adequate accountability of all used and unused study drug. This includes acknowledgement of receipt of each shipment of study drug (quantity and condition), subject administration and dispensing records, and returned or destroyed study product. Administration and dispensing records will document quantities received from Gilead Sciences and quantities administered/dispensed to subjects, including the lot number, date administered/dispensed, subject identification number, subject initials, and the initials of the person dispensing the medication. All used and unused study drug administered/dispensed to subjects must be returned to the site.

Investigational Drug Accountability records will be provided to each study site to:

- Record the date and quantity of study drug received
- Record the date, subject number, subject initials, and the study drug assigned
- Record the date, quantity of used and unused study drug. Dispensing records will include the initials of the person recording the information.

# 5.6.1. Investigational Medicinal Product Return or Disposal

At the start of the study, the study monitor will evaluate each study center's study drug disposal procedures and provide appropriate instruction for return or destruction of unused study drug supplies. If the site has an appropriate Standard Operating Procedure (SOP) for drug destruction, the site may destroy used (empty bottles) and unused study drug supplies performed in accordance with the site's (hospital/pharmacy) SOP. If the site does not have acceptable procedures in place for drug destruction, arrangements will be made between the site and Gilead Sciences (or Gilead Sciences' representative) for return of unused study drug supplies. A copy of the site's SOP will be obtained for central files. Where possible, study drug will be destroyed at the site. Upon study completion, a copy of the Investigational Drug Accountability records must be filed at the site. Another copy will be returned to Gilead Sciences. If drug is destroyed on site, the investigator must maintain accurate records for all study drug bottles destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and person who disposed of the drug. All study drug records must be maintained at the site and copies must be submitted to Gilead Sciences at the end of the study.

## 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows.

The site must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

## 6.1. Subject Enrollment and Treatment Assignment

It is the responsibility of the investigator to ensure that subjects are eligible to participate in the study prior to enrollment and throughout the study.

Documentation of the personally signed and dated informed consent of each subject, using the study-specific ICF, is required before initiating the Screening process. In subjects with HE, which may impair decision-making, consent will be obtained per hospital procedures (eg, by Legally Authorized Representative).

After written informed consent has been obtained and eligibility to participate established, investigative site personnel will obtain the subject's identification number and study drug assignment from the IWRS.

#### 6.2. Pretreatment Assessments

## **6.2.1.** Screening Visit

Local laboratory results obtained within one day of Screening may be used to determine eligibility.

Chest x-rays, local laboratory testing for Hepatitis B and C and HIV Serology, and urine drug testing done during the current hospitalization (which includes transfers from other institutions) and within 10 days of Screening may be used to determine eligibility. A urine pregnancy test must be done locally on the day of the Screening visit.

# <u>NOTE:</u> All subjects will require an additional set of Screening labs drawn for central lab processing.

Subjects will be screened within 14 days prior to randomization to determine eligibility for participation in the study.

The interval between hospitalization and Baseline/Day 1 must be  $\leq$  14 days. This window may be extended under special circumstances with explicit approval from the Medical Monitor.

Subjects who fail to meet eligibility criteria due to an abnormal laboratory result may undergo re-testing of the abnormal analyte once during the Screening window.

Upon pre-approval by the Medical Monitor, subjects who fail to meet eligibility criteria may be re-screened once if there is a reasonable expectation that the subject will meet eligibility after repeat screening.

## Day -14 to Day 0

The following will be performed and documented at Screening:

- Obtain written informed consent
- PPD
- Obtain medical history
- Review and record whether the subject has met inclusion/exclusion criteria
- AUDIT / SADQ questionnaire
- Assess alcohol consumption
- Complete PE including, vital signs, body weight, and height
- Record all concomitant medications that the subject has taken within 30 days prior to Screening
- Perform standard 12-lead ECG
- The following laboratory tests will be collected and performed at **<u>both</u>** the local and central laboratories:
  - Urine sample for drug screen
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatinine, glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, gamma-glutamyl transferase (GGT)
  - Coagulation Tests: PT, PTT, and INR
  - HBsAg
  - Anti-HCV with HCV RNA reflex if positive antibody
  - HIV antibody

Note: Eligibility will be based on local laboratory results.

However, subjects whose HIV or hepatitis B or C serologies from the central laboratory are positive must stop study drug within 3 days of receipt of results. All subjects stopping study drug for these reasons should attend an EoT visit as soon as possible and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study.

The following tests will be performed by the local laboratory **only**:

- Urine samples for urinalysis (routine and microscopic) and culture
- Urine Pregnancy Test (only for female subjects of childbearing potential)
- Blood cultures

Note: Subjects may be eligible based on their local urine pregnancy test; however, if the subject has a positive serum pregnancy test from central laboratory testing (see below), the subject must stop study drug immediately upon receipt of the central laboratory result, attend an EoT visit as soon as possible, and have a follow-up visit 30 days after their last dose of study drug, prior to being withdrawn from the study.

- Obtain blood samples for the following to be sent to the central laboratory **only**:
  - Blood for Biomarkers
  - Insulin
  - Lipid Profile
  - Serum Pregnancy Test (only for females subjects of childbearing potential)
- Assessments for HE, ascites, Hepatorenal Syndrome (HRS), and infection
- Perform chest x-ray (posteroanterior [PA] film is mandatory and a lateral film should be performed if feasible). Chest x-rays performed during the current hospitalization (which includes transfers from other institutions) and within 10 days of Screening are acceptable.
- Perform liver ultrasound (it is acceptable to use a liver ultrasound previously performed during the current hospitalization, including transfers between hospitals.)
- Perform paracentesis (ascitic fluid tap) with ascitic fluid cell count, differential, and culture if clinically-detectable ascites is present (laboratory specimens to be analyzed by the local laboratory only)

## • Perform liver biopsy

Note: Can be performed up to 7 days post Baseline/Day 1. Liver biopsy obtained during the current hospitalization (including transfers between hospitals) prior to Screening is acceptable. However, if biopsy results are not consistent with AH, the subject will stop study drug within 3 days of receipt of the liver biopsy result, attend an EoT visit as soon as possible, and have a follow-up visit 30 days after their last dose of study drug, prior to being withdrawn from the study. If the liver biopsy sample is inadequate to confirm a pathologic diagnosis of AH and no alternative diagnosis is suggested on biopsy, then the subject may remain in the study.

• Record any serious adverse events (SAEs) and all adverse events related to protocol-mandated procedures occurring after signing of the consent form

From the time of obtaining informed consent through the first administration of investigational medicinal product, record all SAEs, as well as any adverse events related to protocol-mandated procedures on the adverse events case report form (eCRF). All other untoward medical occurrences observed during the Screening period, including exacerbation or changes in medical history are to be captured on the medical history eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

Subjects must meet all of the inclusion criteria and none of the exclusion criteria prior to randomization into the study.

## 6.2.2. Baseline / Day 1 Assessments and Randomization

After review of inclusion and exclusion criteria to confirm eligibility, subjects will be randomized to study drug assignment and receive their Subject Identification Number via the IWRS prior to their first dose of study drug.

Randomization will be stratified by MELD < or  $\ge 25$  at Screening as calculated using local laboratory tests and an online MELD calculator (see Section 6.9.7).

During the entire hospitalization period, subjects will be evaluated daily with assessments to include a review of adverse events, concomitant medications, study drug adherence, and a symptom-directed PE including assessments for ascites and HE. Findings based on these assessments and laboratory investigations obtained by treating physicians as part of routine care will be assessed by the investigator for triggers that may necessitate further evaluation and/or treatment discontinuation and managed accordingly per Section 7.5 of the protocol.

The following will be performed and documented at the randomization visit prior to dosing:

- Review inclusion/exclusion criteria and confirm eligibility
- QoL Questionnaire (CLDQ)

- Assess alcohol consumption
- Complete PE including vital signs and body weight
- Perform standard 12-lead ECG
- Assessments for HE, ascites, HRS, and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT. Samples should be drawn for central and local laboratory testing for the calculation of the Lille Score (Section 6.9.12)
  - Coagulation Tests: PT, PTT, and INR. Samples should be drawn for central and local laboratory testing for calculation of the Lille Score (Section 6.9.12)
  - Blood and Urine for Biomarkers
  - ELF<sup>TM</sup> Test and LOXL2
  - Insulin
  - Hemoglobin Alc
  - Lipid Profile
  - Sparse PK Sample (collected after dosing)
  - PPD
- Urine pregnancy test (for females of childbearing potential)
- Collect stool for microbiome testing
- Record all concomitant medications that the subject has taken since the previous visit
- Record any SAEs and all adverse events occurring after signing of the consent form
- Randomization via IWRS (Note: stratification assignment is based on MELD score as calculated using local laboratory results and an online MELD calculator (see Section 6.9.7).

- Administer or dispense GS-4997/placebo and prednisolone, and provide subject with dosing instruction on appropriate dosing and administration
- FibroScan (if available and for subjects without ascites).

#### 6.3. Treatment Assessments

## 6.3.1. Week 1 Visit (±3 Days)

During the Week 1 safety visit the following will be performed and documented:

- Review of liver biopsy and central laboratory results if unavailable during the Screening or baseline period and reassess study entry criteria.
- Assess alcohol consumption
- Complete PE including, vital signs
- Assessments for HE, ascites, HRS, and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT. Samples should be drawn for central and local laboratory testing for calculation of the Lille Score (Section 6.9.12)
  - Coagulation Tests: PT, PTT, and INR.
  - Blood for Biomarkers
  - Sparse PK Sample
- Record all concomitant medications that the subject has taken since the previous visit
- Record any SAEs and all adverse events occurring since the previous visit
- Administer or dispense prednisolone, and provide subject with dosing instruction on appropriate dosing and administration.
- PPD
- Assess for study drug adherence

- Perform study drug accountability
- Calculate Lille Score at Week 1 based on local laboratory results (Section 6.9.12). If Lille score is ≥ 0.56 (null response), prednisolone treatment should be held. If Lille score is > 0.85, then both study drugs should be held. If the central lab results confirm Lille score stopping criteria has been met, the subject will be prematurely discontinued from study drug(s), as appropriate.

# 6.3.2. Week 2 Visit (±3 Days)

During the Week 2 safety visit, the following will be performed and documented:

- Assess alcohol consumption
- Complete PE including vital signs
- Assessments for HE, ascites, HRS and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT. Samples should be drawn for central and local laboratory testing for the calculation of the Lille Score (Section 6.9.12)
  - Coagulation Tests: PT, PTT, and INR
  - Blood for Biomarkers
  - Sparse PK Sample
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit
- PPD
- Assess for Study Drug adherence
- Perform study drug accountability
- Calculate Lille Score at Week 2 based on local laboratory results (Section 6.9.12). If Lille score is > 0.85, then both study drugs should be held. If the central lab results confirm Lille

score stopping criteria have been met, the subject will be prematurely discontinued from study drug(s), as appropriate.

# 6.3.3. Week 3 Visit (±3 Days)

During the Week 3 safety visit, the following will be performed and documented:

- Assess alcohol consumption
- Complete PE including vital signs
- Assessments for HE, ascites, HRS and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT. Samples should be drawn for central and local laboratory testing for the calculation of the Lille Score (Section 6.9.12)
  - Coagulation Tests: PT, PTT, and INR
- Record all concomitant medications that the subject has taken since the previous visit
- Record any SAEs and all adverse events occurring since the previous visit
- Administer or dispense prednisolone, and provide subject with dosing instruction on appropriate dosing and administration
- PPD
- Assess for study drug adherence
- Perform study drug accountability
- Calculate Lille Score at Week 3 based on local laboratory results (Section 6.9.12). If Lille score is > 0.85, then both study drugs should be held. If the central lab results confirm Lille score stopping criteria have been met, the subject will be prematurely discontinued from study drug(s), as appropriate.

# 6.3.4. Week 4 / End of Treatment Visit (EoT) (±3 days)

If the subject meets criteria for discontinuation of treatment (see Section 6.8 of this protocol), the subject should complete an EoT visit as soon as possible after all study drugs are discontinued and attend post-treatment visits as outlined in Appendix 2. Subjects discontinued prior to Week 2 should attend a 30-day FU visit to collect safety data within 30 days of their last dose of study drug. Subjects that have their scheduled Week 4/End of Treatment visit prior to Day 28 will require a phone contact between Study Days 28-35 to assess mortality and liver transplantation.

Subjects should be instructed <u>not to take</u> study drug in the morning of the Week 4 Visit. The dose should be taken as soon as possible after the trough PK (Sparse PK sample collected prior to dosing) and biomarker assessments are completed.

The following will be performed and documented at this visit:

- QoL Questionnaire (CLDQ)
- Assess alcohol consumption
- Complete PE including, vital signs, and body weight
- Perform standard 12-lead ECG
- Assessments for HE, ascites, HRS, and infection.
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT. Samples should be drawn for central and local laboratory testing for the calculation of the Lille Score (Section 6.9.12)
  - Coagulation Tests: PT, PTT, and INR
  - Blood and Urine for Biomarkers
  - ELF<sup>TM</sup> Test and LOXL2
  - Insulin
  - Lipid Profile
  - Sparse PK Sample

- Urine pregnancy test (for females of childbearing potential)
- Collect stool for microbiome testing
- Record all concomitant medications that the subject has taken since the previous visit
- Record any SAEs and all adverse events occurring since the previous visit
- Assess for study drug adherence
- Perform study drug accountability
- FibroScan (if available and for subjects without ascites)
- Record local laboratory results for total bilirubin so that Lille score can be calculated using local laboratory data.

# 6.3.5. Follow Up Visit (±5 Days)

Subjects should return for a Follow-Up Visit 30 days after their last dose of study drug.

Subjects whose liver biopsy results are not consistent with AH or whose HIV or hepatitis B or C serologies from the central laboratory are positive, must stop study drug within 3 days of receipt of results. If the liver biopsy sample is inadequate for pathologic diagnosis of AH and no alternative diagnosis is suggested on biopsy, then the subject may remain in the study. Subjects whose serum pregnancy testing from the central laboratory is positive at Screening must stop study drug immediately upon receipt of this result. All subjects stopping study drug for these reasons should attend an EoT visit as soon as possible and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study. Subjects discontinuing both study drugs prior to Week 2 should complete an end of treatment visit after stopping drug, a 30-day safety FU visit, and all post-treatment follow-up visits. Subjects discontinued after Week 2 should complete an end of treatment assessments as outlined in Appendix 2.

- Record all concomitant medications that the subject has taken since the previous visit
- Record any SAEs and all adverse events occurring since the previous visit
- Assessments for HE, ascites, HRS and infection

- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT
  - Coagulation Tests: PT, PTT, and INR

#### 6.4. Pharmacokinetic Assessments

## 6.4.1. Sparse PK

Blood samples for PK assessments will be collected for all subjects on Baseline/Day 1 and Weeks 1, 2, and 4.

- Baseline/Day 1 sample should be collected  $2 (\pm 1)$  hrs postdose.
- Weeks 1 and 4 samples should be collected at 24 (±4) hrs after previous dose (prior to dosing on visit day). Subjects should not dose until the PK sample is collected.
- Week 2 samples should be collected at 24 (±4) hrs after prior dose (prior to dosing on visit day) AND at 2 (±1) hrs postdose. Subjects should dose in office after the first PK sample is collected.

If a subject requires hemodialysis/hemoperfusion/peritoneal/CRRT dialysis therapy, additional PK samples will be collected on a single occasion during the 4 week treatment period as described below. The start and stop date and time of dialysis, the type of dialysis, and, where applicable, the flow rate of dialysate, will be recorded.

If a subject requires hemodialysis/hemoperfusion/peritoneal dialysis therapy, PK samples should be collected at any single session at the following timepoints:

- Within 30 minutes prior to initiation of the procedure (0 hr)
- Where possible, a single sample from arterial side and a single sample from venous side of the dialyzer approximately 1 hr prior to conclusion of dialysis
- Upon completion of the procedure (within 15 minutes)
- Approximately 1 hr after completion of the procedure.

If a subject requires continuous renal replacement therapy (CRRT), PK samples should be collected on a single occasion any time after the subject has started CRRT at the following timepoints:

- First PK sample: ≥ 6 hours postdose
- Where possible, a single sample from arterial side and a single sample from venous side of the dialyzer approximately 2 hours after first PK sample
- Approximately 3 hours after first PK sample
- Approximately 4 hours after first PK sample

Note: If a subject discontinues treatment, but remains in the study, PK samples do not need to be collected after the end of treatment visit.

## 6.4.2. Intensive PK Substudy

PPD

#### 6.5. Post-Treatment Assessments

### 6.5.1. Week 6 ( $\pm$ 3 Days)

Subjects will return for Follow-Up Visits starting at Week 6 after the Week 4 / EoT Visit or the last dose of study drug to undergo the following:

- Assess alcohol consumption
- Complete PE including vital signs
- Assessments for HE, ascites, HRS and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT
  - Coagulation Tests: PT, PTT, and INR.

- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

## 6.5.2. Weeks 8, 16, and 20 / Post Treatment Visits ( $\pm$ 5 Days)

During the Week 8, 16, and 20 post treatment visits, the following will be performed and documented:

- Assess alcohol consumption
- Complete PE including, vital signs
- Perform standard 12-lead ECG (Week 8 only)
- Assessments for HE, ascites, HRS and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT
  - Coagulation Tests: PT, PTT, and INR
  - Blood for Biomarkers (Week 8 only)
- Urine pregnancy test (for females of childbearing potential)
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit (Week 8 only)
- Record procedure-related adverse events and procedure-related SAEs as well as any SAEs that the investigator deems relevant to the use of study drug for Weeks 16 and 20 only
- Subjects that have their scheduled Week 8 visit prior to Day 56 will require a phone contact between Day 56-63 respectively, to assess for mortality and liver transplantation.

# 6.5.3. Weeks 12 and 24 / Post Treatment Visits (± 5 Days)

Subjects that have their scheduled Week 12 or Week 24 visit prior to Day 84 or Day 168, will require a phone contact between Day 84-91 or Day 168-175 respectively, to assess for mortality and liver transplantation.

During the Week 12 and Week 24 post treatment visits, the following will be performed and documented:

- QoL Questionnaire (CLDQ, week 24 only)
- Assess alcohol consumption
- Assessments for HE, ascites, HRS and infection
- Complete PE including, vital signs, and body weight
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT
  - Coagulation Tests: PT, PTT, and INR
  - Blood for Biomarkers; Urine for Biomarkers (Week 24 only)
  - ELF<sup>TM</sup> Test and LOXL2
  - Insulin
  - Hemoglobin A1c
  - Lipid Profile
- Stool for microbiome testing (week 24 only)
- Urine pregnancy test (for females of childbearing potential)
- Record all concomitant medications that the subject has taken since the previous visit
- Record all serious adverse events and any study related adverse events occurring since the previous visit

- Record procedure-related adverse events and procedure-related SAEs as well as any SAEs that the investigator deems relevant to the use of study drug (Week 24 only)
- FibroScan (if available and for subjects without ascites [Week 24 only])

#### 6.6. Unscheduled Visits

Additional unscheduled assessments may be performed at the discretion of the investigator. At a minimum, the following will be performed and documented, unless the unscheduled visit is only to refill medication, then the following procedures are not necessary.

- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit
- Assessments for HE, ascites, HRS and infection
- Obtain blood samples for:
  - Hematology
  - Chemistry: ALT, AST, albumin, alkaline phosphatase, bicarbonate, BUN, calcium, chloride, creatinine, glucose, LDH, magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, GGT
  - Coagulation Tests: PT, PTT, and INR

## 6.7. Assessments for Premature Discontinuation from Study

Discontinuation from study drug dosing and discontinuation from the study (including follow-up visits and phone contact at Week 8, Week 12, and Week 24) are 2 distinct actions.

Subjects with histologically confirmed AH who discontinue study drug (for any reason other than death) prior to completion of the assigned dosing period, should complete an EoT visit, a 30 day follow up visit, and all required follow-up study visits.

Subjects whose liver biopsy results are not consistent with AH or whose HIV or hepatitis B or C serologies from the central laboratory are positive, must stop study drug within 3 days of receipt of results. Subjects whose serum pregnancy testing from the central laboratory is positive at Screening must stop study drug immediately upon receipt of this result. All subjects stopping study drug for these reasons should attend an EoT visit as soon as possible and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study. These subjects will not complete the remaining follow-up study visits.

Subjects are considered to have completed the study after the Follow up Week 24 visit, regardless of treatment duration and/or early termination from study drug.

# 6.8. Criteria for Discontinuation of Study Treatment

Study medication must be discontinued in the following instances:

- Liver biopsy inconsistent with diagnosis of AH. If the liver biopsy sample is inadequate for pathologic diagnosis of AH and no alternative diagnosis is suggested on biopsy, then the subject may remain in the study.
- Serologies for HIV, hepatitis B, or hepatitis C from central laboratory testing are positive
- Serum pregnancy test at Screening from central laboratory testing is positive, and /or pregnancy during the study; refer to Appendix 3
- Subject who develops a SAE consisting of a serious allergic reaction to the study drug
- Unacceptable toxicity, or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific procedures or is considered to not be in the subject's best interest
- Subject request to discontinue for any reason
- Discontinuation of the study at the request of Gilead, a regulatory agency or an institutional review board or independent ethics committee (IRB/IEC/EC)

Study medication may be discontinued with discretion in the following instances:

- Intercurrent illness that would, in the judgment of the investigator, affect assessments of clinical status to a significant degree. Following resolution of intercurrent illness, the subject may resume study dosing at the discretion of the investigator after discussion with the Medical Monitor
- Potential drug-related hepatotoxicity; refer to Section 7.5
- Subject noncompliance
- Sponsor discretion

# 6.9. Description of Assessments

## 6.9.1. Liver Biopsy

A core liver biopsy via either the percutaneous or transjugular route will be performed at Screening. Liver biopsy obtained during the current hospitalization (including transfers between hospitals) prior to Screening is acceptable. Liver biopsy can be performed up to 7 days following the Baseline/Day 1 visit. Subjects may start treatment prior to receipt of the liver biopsy result if the subject has met all other eligibility criteria. In such cases, if a diagnosis consistent with AH is not confirmed on the liver biopsy, the subject must stop study drugs within 3 days of receipt of the liver biopsy result, attend an EoT visit as soon as possible, and have a follow-up visit 30 days after their last dose of study drug, prior to being withdrawn from the study. At minimum, a histological diagnosis of AH consists of the presence of hepatocellular injury characterized by hepatocyte ballooning, neutrophilic infiltration, and steatosis {Lucey 2009}. Grading of liver biopsies according to the Alcoholic Hepatitis Histologic Score (AHHS) is preferred {Angeli 2015}. If the liver biopsy sample is inadequate for a pathologic diagnosis of AH, but does not reveal another etiology, the subject may remain in the study.

# 6.9.2. Electrocardiogram

Standard 12-lead electrocardiogram (ECG) assessments will be performed. The Investigator will review the ECGs for any clinically significant abnormalities to ensure subject safety. Abnormal ECG findings that are considered clinically significant by the Investigator and meet the definition of an AE should be reported and recorded on the AE case report form.

## **6.9.3. AUDIT / SADQ Questionnaires**

The Alcohol Use Disorders Identification Test (AUDIT) is a 10-question test to determine if the subject may be at risk for alcohol abuse problems.

The Severity of Alcohol Dependence Questionnaire (SADQ) is a 20-question test to measure the presence of alcohol dependence.

AUDIT and SADQ will be completed by subjects at the Screening visit. A Legally Authorized Representative may assist the subject in completing the questionnaires. It is recommended to administer these questionnaires prior to the clinical and laboratory assessments. If the subject is unable or refuses to complete a questionnaire, this should be documented on the relevant eCRF.

## 6.9.4. Quality of Life (QoL) Measures

The Chronic Liver Disease Questionnaire (CLDQ) will be collected at Baseline/Day 1, Week 4, and Week 24. It is recommended to administer this questionnaire prior to the clinical and laboratory assessments. Legally Authorized Representative may assist the subject in completing the questionnaires. If the subject is unable or refuses to complete a questionnaire, this should be documented on the relevant eCRF. The CLDQ asks 29 questions related to liver disease to measure health related quality of life in subjects with chronic liver disease.

## 6.9.5. Hepatic Encephalopathy (HE)

The severity of HE should be graded according to the West Haven Criteria, which are based on changes of consciousness, intellectual function, and behavior.

- Grade 1 Trivial lack of awareness; euphoria or anxiety; shortened attention span; impaired performance of addition
- Grade 2 Lethargy or apathy; minimal disorientation for time or place; subtle personality change; inappropriate behavior; impaired performance of subtraction
- Grade 3 Somnolence to semistupor, but responsive to verbal stimuli; confusion; gross disorientation
- Grade 4 Coma (unresponsive to verbal or noxious stimuli)

Medications used to treat HE should be recorded on the concomitant medications case report form.

#### **6.9.6.** Ascites

The severity of ascites should be graded according to the following modification of the International Ascites Club Criteria.

- Grade 0 No ascites detectable clinically or by ultrasound
- Grade 1 Mild ascites only detectable by ultrasound
- Grade 2 Moderate ascites evident by moderate symmetrical distension of abdomen
- Grade 3 Large or gross ascites with marked abdominal distension

Medications used to treat ascites should be recorded on the concomitant medications case report form. If a subject has Grade 0 or 1 ascites, but is taking diuretic therapy for treatment, record ascites as Grade 2.

## 6.9.7. Maddrey's DF, MELD and Child-Pugh-Turcotte Scores

For purposes of inclusion/exclusion criteria, local laboratory results and online calculators will be used to calculate the Maddrey's DF and MELD scores at Screening. Specifically, Maddrey's DF will be calculated at the Screening visit based on local laboratory results for PT, PT control, and serum total bilirubin. The following online calculator will be used: http://www.gastrotraining.com/calculators/maddreys-discriminant.

The screening MELD score will be calculated based on the local laboratory results for INR, serum creatinine, and total bilirubin in appropriate units (SI or conventional) at the Screening

visit using the following online calculator: http://www.mdcalc.com/original-meld-score-pre-2016-model-for-end-stage-liver-disease.

# <u>NOTE:</u> The MELD online calculator uses the original pre-2016 MELD formula without the adjustment for Sodium.

MELD score, Child-Pugh-Turcotte (CPT) score, and Maddrey's DF will be assessed at each study visit (see Appendix 4 for more information regarding the CPT scoring and classification). Components of the MELD, CPT, and Maddrey's DF scores which are based on laboratory values, the data will be obtained from the central laboratory within the clinical database for analysis.

## 6.9.8. Hepatorenal Syndrome (HRS)

The occurrence of HRS should be confirmed based on the following diagnostic criteria from the International Ascites Club (IAC) {Angeli 2015}. The date of diagnosis/resolution and specific therapies for HRS should be recorded.

- Cirrhosis with ascites
- Diagnosis of acute kidney injury (AKI) according to the ICA-AKI criteria
  - Definition of AKI: Increase in serum creatinine  $\geq 0.3$  mg/dL ( $\geq 26.5$  µmol/L) within 48 hours or a percentage increase of  $\geq 50\%$  from Baseline/Day 1.
  - Stages:
    - 1: Increase in serum creatinine  $\geq 0.3$  mg/dL ( $\geq 26.5$  µmol/L) or an increase  $\geq 1.5x$  to 2x from Baseline/Day 1.
    - 2: Increase in serum creatinine > 2-3x from Baseline/Day 1.
    - 3: Increase in serum creatinine > 3x from Baseline/Day 1 or serum creatinine  $\geq 4.0 \text{ mg/dL}$  ( $353.6 \mu \text{mol/L}$ ) with an acute increase  $\geq 0.3 \text{ mg/dL}$  ( $\geq 26.5 \mu \text{mol/L}$ ) from Baseline/Day 1 or initiation of renal replacement therapy.
  - Stage 2 or 3 AKI without improvement of serum creatinine to stage 1 AKI after at least 2 days with diuretic withdrawal and volume expansion with albumin. The recommended dose of albumin is 1 g/kg of body weight per day up to a maximum of 100 g/day.
- Absence of shock
- No current or recent treatment with nephrotoxic drugs

• Absence of parenchymal renal disease as indicated by proteinuria >500 mg/day, microhematuria (> 50 red blood cells per high power field) and/or abnormal renal ultrasonography.

After the diagnosis of HRS, treatment with vasoconstrictors and albumin is recommended. Where available, terlipressin is recommended based on the EASL Clinical Practice Guidelines (http://www.easl.eu/research/our-contributions/clinical-practice-guidelines/detail/management-of-ascites-spontaneous-bacterial-peritonitis-and-hepatorenal-syndrome-in-cirrhosis/report/6); norepinephrine or midodrine plus octreotide are acceptable alternatives based on AASLD Practice Guidelines

 $(http://www.aasld.org/sites/default/files/guideline\_documents/adultascitesen hanced.pdf).\\$ 

### 6.9.9. Infection

The occurrence of bacterial, fungal, or viral infections should be recorded as adverse events. Relevant data to be recorded include the source of infection, date of onset/resolution, presence of fever (temperature ≥ 38°C/100.4°F), laboratory investigations (e.g. white blood cell count, cultures, chest x-ray), and anti-microbial therapy. An infection will be considered definite in subjects with clinical evidence of infection and a positive culture from a normally sterile source (with the exception of spontaneous bacterial peritonitis [SBP] as below). All other infections will be considered probable. In subjects with ascitic fluid neutrophils ≥ 250 cells/mm³, definite SBP will be recorded irrespective of culture positivity.

If pneumonia develops during the study, treatment according to the following guidelines is recommended:

- Community-Acquired Pneumonia: Infectious Diseases Society of America/American Thoracic Society Consensus Guidelines (2007) (http://cid.oxfordjournals.org/content/44/Supplement\_2/S27.full)
  - The minimum recommended duration of antibiotic treatment is 5 days.
- Hospital-Acquired Pneumonia (HAP): Infectious Diseases Society of America/American
  Thoracic Society Consensus Guidelines (2016)
  (http://www.idsociety.org/Guidelines/Patient\_Care/IDSA\_Practice\_Guidelines/Infections\_by
  \_Organ\_System/Lower/Upper\_Respiratory/Hospital-Acquired\_Pneumonia\_(HAP)/)
  - HAP is defined as a pneumonia not incubating at the time of hospital admission and occurring ≥ 48 hours after admission.
  - The minimum recommended duration of antibiotic treatment is 7 days.

SBP, UTI, and other infections that develop during the study should be treated according to the following guidelines:

- SBP: AASLD Practice Guidelines: Management of Adult Patients with Ascites Due to Cirrhosis: Update 2012. (http://www.aasld.org/publications/practice-guidelines-0#practice\_guidelines\_accordion-block-2). The minimum recommended duration of antibiotic treatment is 5 days. Patients with SBP who also have a serum creatinine > 1 mg/dL, blood urea nitrogen > 30 mg/dL, or total bilirubin > 4 mg/dL should also receive 1.5 g albumin per kg body weight within 6 hours of detection and 1.0 g/kg 2 days later.
- UTI: American Urological Association Adult UTI Guidelines (2016) (https://www.auanet.org/education/adult-uti.cfm). The minimum recommended duration of antibiotic treatment is 5 days for uncomplicated UTI, 7 days for uncomplicated UTI in patients with diabetes, and 14 days for complicated UTI.
- Other infections: Investigator's discretion.

In subjects with documented infection, interruption of prednisolone should be considered at the discretion of the investigator (see Section 7.5: Toxicity Management). GS-4997/placebo does not require dose modification in subjects with infection.

## 6.9.10. Screening Laboratory Assessments

All samples for laboratory assessments will be sent to the central laboratory with the exception of urine samples for urinalysis and culture, blood cultures and urine pregnancy tests which will be completed at the site.

The following laboratory tests will be collected at Screening for testing at both the local and central laboratories: urine drug screen, hematology, chemistry, coagulation tests, hepatitis B serology, hepatitis C serology, and HIV serology.

Chest-x-rays and local laboratory testing for Hepatitis B and C and HIV Serology and urine drug testing done during the current hospitalization (which includes transfers from other institutions) and within 10 days of Screening may be used to determine eligibility. A urine pregnancy test must be done locally on the day of the Screening visit. An additional set of Screening labs must be drawn for central laboratory processing.

However, for hepatitis B serology, hepatitis C serology, and HIV serology, eligibility is confirmed based on central laboratory testing. Subjects may be enrolled based on local urine pregnancy testing, but serum pregnancy testing via the central laboratory will be the basis for final eligibility to continue the subject in the study. Refer to Section 6.7 for assessments to be completed for premature discontinuation from the study.

Specific instructions for processing, labelling, and shipping samples will be provided in a central laboratory manual.

# 6.9.11. FibroScan®

Where available, liver stiffness measurement by FibroScan® will be performed at Baseline/Day 1, Week 4 and Week 24. Liver stiffness measurement should not be performed in subjects with ascites. At each visit, median liver stiffness (in kilopascals (kPa)), and where available, the median Controlled Attenuation Parameter (CAP) value will be recorded.

#### 6.9.12. Lille Score

The Lille score should be calculated at Day 7 using local laboratory results from Baseline/Day 1 (albumin, total bilirubin, creatinine, PT) and Week 1 (total bilirubin) for all subjects utilizing the following calculator (http://www.mdcalc.com/lille-model-alcoholic-hepatitis/), in appropriate units (SI or conventional).

Prednisolone should be discontinued in subjects with a Lille Score  $\geq 0.56$  at Day 7 (null response); these subjects may continue GS-4997/placebo treatment.

For safety monitoring of the stopping criteria of Lille score > 0.85, sites should also collect local laboratory results for total bilirubin at Weeks 2, 3, and 4 and use the same calculator to calculate the Lille Score compared to baseline values. When performing the calculation, ensure the Day 7 total bilirubin is changed to Week 2, 3, and 4 values at the appropriate time points.

If a subject's Lille score is > 0.85 at any time, they should stop both study drugs. If the central laboratory Lille score calculation is different from the local laboratory results, the stopping criteria will be based on central laboratory results.

# **6.10.** End of Study Definition

The end of the study will be the last subject's last observation (or visit).

## 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post-treatment complications that occur as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the Screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (eg, hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history CRF.

### 7.1.2. Serious Adverse Events

A **serious adverse event** (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization

- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

# 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to IMP therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the IMP. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the investigational medicinal product.
It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures, (eg, venipuncture)

## 7.2.2. Assessment of Severity

The severity grading of AEs will be assessed as Grade 1, 2, 3, or 4 according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, which can be found at http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE 4.03 2010-06-14 QuickReference 5x7.pdf.

For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

The distinction between the seriousness and the severity of an adverse event should be noted. Severe is a measure of intensity; thus, a severe reaction is not necessarily a serious reaction. For example, a headache may be severe in intensity, but would not be classified as serious unless it met one of the criteria for serious events listed above.

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead

Requirements for collection prior to study drug initiation:

After informed consent, but prior to initiation of study medication, the following types of events should be reported on the case report form (eCRF): all SAEs and adverse events related to protocol-mandated procedures.

#### **Adverse Events**

Following initiation of study medication, collect all AEs, regardless of cause or relationship, until 30 days after last administration of study IMP must be reported to the eCRF database as instructed. During the post-treatment follow-up period (through Week 24), AEs including SAEs related to protocol mandated procedures must be collected and reported to the eCRF database.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the protocol defined follow up period.

#### **Serious Adverse Events**

All SAEs including deaths, regardless of cause or relationship, that occurs after the subject first consents to participate in the study (ie, signing the informed consent) until 30days after the last dose of study IMP must be reported to the eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This also includes any SAEs resulting from protocol-associated procedures performed after informed consent is signed. During the post-treatment follow-up period (through Week 24) any SAEs deemed related to the use of study IMP should also be reported.

Investigators are not obligated to actively seek SAEs after the protocol defined follow up period. However, if the investigator learns of any SAEs that occured after study participation has concluded and the event is deemed relevant to the use of IMP, he/she should promptly document and report the event to Gilead DSPH.

- All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guideline.
- Electronic Serious Adverse Event (eSAE) Reporting Process
- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours to:

Gilead Sciences DSPH Fax: +1 (650) 522-5477

E-mail: Safety FC@gilead.com

- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other documents are also to be submitted by e-mail or fax when requested and applicable. Transmission of such documents should occur without personal subject identification, maintaining the traceability of a document to the subject identifiers.

- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the event description section of the SAE form.

## 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study IMP. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

## 7.5. Toxicity Management

Treatment-emergent toxicities will be noted by the Investigator and brought to the attention of the Medical Monitor. Whether or not considered treatment-related, all subjects experiencing AEs must be monitored periodically until symptoms subside, any abnormal laboratory values have resolved or returned to baseline levels or they are considered irreversible, or until there is a satisfactory explanation for the changes observed.

Administration of all study drugs may be discontinued due to a clinical or laboratory adverse event. Subjects are allowed to take one study drug and not the other.

Prednisolone may be dose-reduced or interrupted at the discretion of the investigator (e.g. due to new-onset, severe sepsis or diabetes mellitus that cannot adequately be controlled). Prednisolone should be discontinued in subjects with a Lille Score ≥ 0.56 at Day 7 (null responders); these subjects may continue GS-4997/placebo treatment. Except in Lille Score null responders, restarting prednisolone may be considered if the reason for interruption has resolved or become adequately controlled in the opinion of the investigator within 7 days of prednisolone interruption. Any decision to restart prednisolone must be reviewed with the Medical Monitor.

There is no option for GS-4997/placebo dose reduction, but GS-4997/placebo may be interrupted due to drug-related toxicity (see below). If GS-4997/placebo is interrupted, it may be restarted on

a case by case basis if the reason for interruption has resolved or become adequately controlled in the opinion of the investigator within 7 days of GS-4997/placebo interruption. Any decision to discontinue or restart GS-4997/placebo must be reviewed with the Medical Monitor.

Subjects who meet any of the following criteria must stop GS-4997/placebo

- Laboratory Criteria (based on central laboratory data):
  - Total bilirubin > 3x Baseline/Day 1 or nadir (confirmed by immediate repeat testing)
  - ALT and/or AST > 5x Baseline/Day 1 (confirmed by immediate repeat testing), unless the elevation is thought by the Principal Investigator to be secondary to an etiology other than GS-4997-related, drug-induced liver injury (e.g. infection).
  - AST and/or ALT >500 U/L should trigger prompt (within 24-48 hours) evaluation of patients for consideration of GS-4997/placebo discontinuation. If patients with AST and/or ALT >500 U/L are continued on study drug, they must be monitored closely with repeat PE and laboratory evaluation at least 3 times per week.
- Lille score > 0.85 at any time point (eg, on/after first scheduled post-Baseline/Day 1 visit) while on study drug (base on central or local laboratory data)
- Any Grade 3 or higher AE assessed as possibly or likely related to GS-4997

Other than in the case of the liver enzymes noted above, Grade 3 or 4 clinically significant laboratory abnormalities should be confirmed by repeat testing as soon as practical to do so (Medical Monitor needs to be notified), and preferably within 3 calendar days of receipt of the original test results.

Clinical events and clinically significant laboratory abnormalities will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, which can be found at http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-14\_QuickReference\_8.5x11.pdf.

When restarting investigational medicinal product following resolution of the adverse event, the investigational medicinal product should be restarted at full dose following discussion with the Medical Monitor.

Any questions regarding toxicity management should be directed to the Medical Monitor.

# 7.5.1. Assessment of Potential Drug-Induced Liver Injury by an Independent Adjudicator

Due to the challenge of recognizing and diagnosing drug-induced liver injury (DILI) in subjects with severe hepatic dysfunction (e.g. due to AH), a hepatologist with expertise in AH and drug-related hepatotoxicity will review potential cases of DILI. Subjects will be categorized as those for whom DILI or worsening of hepatic function (treatment failure) attributable to study

drug could be excluded (e.g. a clear, alternative explanation exists); those for whom DILI or worsening of hepatic function (treatment failure) attributable to study drug could not be excluded (e.g. no clear, alternative explanation exists); and those with insufficient data to make a determination.

The following events will be adjudicated:

- Total bilirubin > 2 × Baseline/Day 1 or nadir and ALT and/or AST > 3 × Baseline/Day 1 or nadir (confirmed by immediate repeat testing)
- Total bilirubin  $> 3 \times Baseline/Day 1$  or nadir (confirmed by immediate repeat testing)
- ALT and/or AST  $> 5 \times$  Baseline/Day 1 (confirmed by immediate repeat testing)
- ALT and/or AST > 500 U/L (confirmed by immediate repeat testing)
- Lille score >0.85 at any time point (eg, on/after first scheduled post-Baseline/Day 1 visit) while on study drug (base on central or local laboratory data)

## 7.6. Special Situations Reports

## 7.6.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, reports of adverse events associated with product complaints, and pregnancy reports regardless of an associated AE.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labelling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

## 7.6.2. Instructions for Reporting Special Situations

## 7.6.2.1. Instructions for Reporting Pregnancies

The investigator should report pregnancies in female study subjects that are identified after initiation of study medication and throughout the study, including the post study drug follow-up period, to Gilead DSPH using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

Refer to Section 7.4 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Sections 7.1.1 and 7.1.2. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead DSPH.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to Gilead DSPH using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety\_FC@gilead.com and Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to Gilead DSPH using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 650 522-5477 or email Safety FC@gilead.com.

Refer to Appendix 3 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

## 7.6.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to Gilead DSPH within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study IMP and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Special situations involving non-Gilead concomitant medications do not need to be reported on the special situations report form; however, for special situations that result in AEs due to a non-Gilead concomitant medication, the AE should be reported on the AE form.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 7.4 and the eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

#### 8. STATISTICAL CONSIDERATIONS

## 8.1. Analysis Objectives and Endpoints

The objectives of the study are described in Section 2 of the protocol, and endpoints for the study are described below.

## 8.1.1. Primary Endpoint

The primary endpoint is the safety of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe AH. Safety and tolerability will be evaluated by examining the incidence of treatment emergent adverse events, including serious adverse events, clinical laboratory tests, ECGs, and vital signs. The number and percentage of subjects who prematurely discontinue study drug due to adverse events will be provided. Adverse events that led to premature study drug discontinuation will be summarized by system organ class and preferred term.

## 8.2. Secondary Endpoints

#### Clinical Outcomes:

- Number (%) of subjects who die by Study Day 28, Week 8, Week 12, and Week 24
- Number (%) of subjects receiving a liver transplant
- Number (%) of subjects with HRS
- Number (%) of subjects with infection
- Length of hospital stay

## Measures of Hepatic Synthetic Function:

- Change from baseline in liver biochemistry tests (ALT, AST, GGT, alkaline phosphatase, bilirubin, albumin and INR) by visit
- Lille response (score < 0.45) at Day 7, Lille null response (score ≥ 0.56) at Day 7, Lille score at Day 7 as a continuous variable, and combined score including Lille score at Day 7 and baseline MELD score
- Change from baseline in prognostic indices (MELD, CPT, and Maddrey's DF scores) by visit





## 8.3. Analysis Conventions

## 8.3.1. Analysis Sets

## 8.3.1.1. Efficacy

The primary analysis set for efficacy analyses will be the Full Analysis Set (FAS) which includes all subjects with histologically-confirmed severe AH who were randomized into the study and received at least one dose of study drug.

Subjects who receive study drug other than that to which they were assigned will be analyzed according to the treatment group to which they were randomized.

## 8.3.1.2. Safety

The primary analysis set for safety analyses will be the Safety Analysis set which includes all subjects who received at least one dose of study drug. Treatment-emergent data will be analyzed and defined as data collected from the first dose of study drug through the date of last dose of study drug plus 30 days. Subjects who received study drug other than that to which they were assigned will be analyzed according to the study drug received.

#### 8.3.1.3. Pharmacokinetics

The Pharmacokinetic (PK) Analysis Set includes all subjects who have been administered at least one dose of active study drug (GS-4997) and have at least one non-missing postdose concentration value for the corresponding analyte in plasma or serum.



## 8.4. Data Handling Conventions

Missing data can have an impact on the interpretation of the trial data. In general, values for missing data will not be imputed.

Where appropriate, safety data for subjects who received study drug but did not complete the study will be included in summary statistics. For example, if a subject received study medication, the subject will be included in a summary of adverse events according to the treatment received; however, if the subject is not dosed then they will be excluded from the summary. If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a predose value, then the subject will be excluded from the calculation of summary statistics for the predose value and the change from predose values.

Values for missing safety laboratory data, ECGs, and vital signs will not be imputed; however, a missing baseline result will be replaced with a Screening result, if available. If no pre-treatment laboratory value is available, the baseline value will be assumed to be normal (ie, no grade [Grade 0]) for the summary of graded laboratory abnormalities.

## 8.5. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods by treatment group. Demographic summaries will include age, sex, race, and ethnicity.

Baseline characteristics summary will include body weight, height, body mass index, baseline MELD, CPT, Maddrey's DF, and other baseline disease characteristic variables of interest.

#### 8.6. Primary Analysis

The primary endpoint is the safety of GS-4997 in combination with prednisolone versus prednisolone alone in subjects with severe AH. The primary analysis will be conducted after all subjects have been followed through 30 days after the date of their last dose of study drug, or been prematurely terminated from study.

## 8.7. Efficacy Analysis

The biological activity of the combination of GS-4997 and prednisolone and prednisolone alone will be evaluated using clinical outcomes (mortality, hepatorenal syndrome [HRS], infection, liver transplantation, and length of hospital stay) and measures of hepatic function (Lille response at Day 7, and change from baseline in MELD, CPT, and Maddrey's DF scores, and liver biochemistry tests).

PPD

The percentage of subjects with Lille score response (defined as a Lille score < 0.45 at Day 7), and percentage of subjects who have died by Day 28 will be compared between treatment groups using a 2-sided Fisher's exact test. Transplantation-free survival to Day 28, Week 8, Week 12 and Week 24 will be analyzed using Kaplan-Meier methods. For continuous variables, an 8-number summary will be provided by treatment group. For categorical variables, descriptive statistics (count and percentage of subjects in each category) will be presented by treatment group. Point estimates (and when appropriate 95% CI) will be calculated for each parameter.

#### 8.7.1. Exploratory Analysis

PPD

#### 8.8. Safety Analysis

Safety will be evaluated by assessment of clinical laboratory tests, PEs, ECGs, and vital signs measurements at various time points during the study, and by the documentation of AEs.

All safety data collected while "on treatment" (ie, on or after the first dose of study drug administration up to 30 days after the last dose of study drug) will be summarized by treatment group according to the study drug received. Safety endpoints will be analyzed as the number and percentage of subjects with events or abnormalities for categorical variables. Continuous

variables will be descriptively summarized (n, mean, standard deviation, median, Q1, Q3, minimum and maximum).

## **8.8.1.** Extent of Exposure

A subject's extent of exposure to study drug will be generated from the study drug administration page of the eCRF. Exposure data will be summarized by treatment group.

#### **8.8.2.** Adverse Events

Clinical and laboratory adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database. Adverse event severity will be graded using the CTCAE Version 4.03.

Events will be summarized on the basis of the date of onset for the event. Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
- Any AEs leading to premature discontinuation of study drug.

Summaries (number and percentage of subjects) of TEAEs by SOC and PT will be provided. Treatment-emergent AEs will also be summarized by relationship to study drug and by severity. In addition, TEAEs leading to premature discontinuation of study drug and study will be summarized and listed

All AEs collected during the course of the study will be presented in data listings with a field for treatment-emergent event (yes/no).

## **8.8.3.** Laboratory Evaluations

Selected laboratory data (using conventional units) will be summarized using only observed data. The value and change from baseline at all scheduled time points will be summarized.

Graded laboratory abnormalities will be defined using the grading scheme in the CTCAE Version 4.03.

Incidence of treatment-emergent grade 3 or higher laboratory abnormalities, defined as most severe grade 3 or higher post-baseline value that has increased by at least one toxicity grade from baseline at any time post baseline up to 30 days after the last dose of study drug, will be summarized by treatment group. If baseline data are missing, then any graded abnormality (ie, at least a Grade 1) will be considered treatment emergent.

## 8.8.4. Other Safety Evaluations

A shift table of the investigator's assessment of ECG results at Week 4/early study drug discontinuation visit and Week 8 compared with baseline values will be presented by treatment group using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant; or missing.

## 8.9. Pharmacokinetic Analysis



## 8.9.1. Other Exploratory Analyses

PPD

## 8.10. Sample Size

The number of subjects was chosen based on clinical experience with other similar proof of concept studies. PPD

## 8.11. Data Monitoring Committee

An independent, external Data Monitoring Committee (DMC) that includes two hepatologists and a PhD statistician will convene prior to study start, once 20 subjects have been treated for 28 days and every 3 months thereafter to monitor the study for safety events including SAEs, death, premature discontinuation of treatment for AEs, Grade 3 and higher AEs, Grade 3 and higher treatment-emergent laboratory abnormalities, and individual subject stopping criteria for GS-4997/placebo study drug (see Section 7.5).

The DMC will also evaluate (based on an unblinded review of safety data) and recommend early termination of the trial if there is a > 20% higher percentage of subjects in the GS-4997/prednisolone group than in the prednisolone alone group with: 1) Grade 3 or higher, treatment-emergent, treatment-related adverse event(s) of a specific type (excluding evaluation of liver function) where GS-4997/Placebo was prematurely withdrawn; 2) death on/prior to Study Day 28; 3) Lille score > 0.85 while on study drug; 4) any of the post-baseline GS-4997/placebo laboratory stopping criteria (ie, ALT or AST > 500 U/L that led to discontinuation of GS-4997/placebo, ALT or AST > 5x Baseline/Day 1 [confirmed on repeat testing]; or total bilirubin > 3 x Baseline/Day 1 or nadir [confirmed on repeat testing]).

The DMC will provide recommendations to Gilead on whether the nature, frequency, and severity of adverse effects associated with study treatment warrant the early termination of the study in the best interest of the participants, whether the study should continue as planned, or the study should continue with modifications. The DMC may also provide recommendations as needed regarding study design.

The DMC's specific activities will be defined by a mutually agreed charter, which will define the DMC's membership, conduct and meeting schedule.

While the DMC will be asked to advise Gilead regarding future conduct of the study, including possible early study termination, Gilead retains final decision-making authority on all aspects of the study.

## 9. **RESPONSIBILITIES**

## 9.1. Investigator Responsibilities

## 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki, International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. These standards are consistent with the European Union Clinical Trials Directive 2001/20/EC and Good Clinical Practice Directive 2005/28/EC.

The investigator will ensure adherence to the basic principles of Good Clinical Practice, as outlined in 21 CFR 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, 1998, and 21 CFR, part 56, 1998.

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, 1998, providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

# 9.1.2. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Ethics Committee (EC) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IRB/IEC/EC. The investigator will not begin any study subject activities until approval from the IRB/IEC/EC and regulatory agency, if required, has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the IRB/IEC/EC for any modifications made to the protocol or any accompanying material to be provided to the subject after initial approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The investigator must use the most current IRB/IEC/EC approved consent form for documenting

written informed consent. Each informed consent (or assent as applicable) will be appropriately signed and dated by the subject or the subject's legally authorized representative and the person conducting the consent discussion, and also by an impartial witness if required by IRB/IEC/EC. The consent form will inform subjects about genomic testing and sample retention, and their right to receive clinically relevant genomic analysis results.

## 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law) and an identification code will be recorded on any form or biological sample submitted to the sponsor, IRB/IEC/EC, or laboratory. Laboratory specimens must be labeled in such a way as to protect subject identity while allowing the results to be recorded to the proper subject. Refer to specific laboratory instructions for further details. NOTE: The investigator must keep a Screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, eCRF, the IMP, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

## 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, CRF and query forms, IRB/IEC/EC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, PE, and confirmation of diagnosis (to support inclusion and exclusion criteria);

- Documentation of the reason(s) a consented subject is not enrolled;
- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of IMP, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

## 9.1.6. Electronic Case Report Forms

For each subject consented, an eCRF will be completed by an authorized study staff member whose training for this function is documented according to study procedures. The eCRF should be completed in a timely manner to enable the sponsor to perform central monitoring of safety data. Subsequent to data entry, a study monitor will perform source data verification within the EDC system. Original entries as well as any changes to data fields will be stored in the audit

trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will use his/her log in credentials to confirm that the forms have been reviewed, and that the entries accurately reflect the information in the source documents. The eCRF capture the data required per the protocol schedule of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (eg, data entry error). At the conclusion of the trial, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5.

## 9.1.7. Investigational Medicinal Product Accountability and Return

The investigator or designee (ie, pharmacist) is responsible for ensuring adequate accountability of all used and unused study drug. This includes acknowledgment of receipt of each shipment of study product (quantity and condition), subject dispensing records, and returned or destroyed study product. Dispensing records will document quantities received from Gilead Sciences and quantities dispensed to subjects, including lot number, date dispensed, subject identifier number, subject initials, and the initials of the person dispensing the medication.

At study initiation, the monitor will evaluate the site's standard operating procedure of investigational medicinal product/destruction in order to ensure that it complies with Gilead Sciences requirements. Drug may be returned or destroyed on an ongoing basis during the study, if appropriate. At the end of the study, following final drug inventory reconciliation by the monitor, the study site will dispose of and/or destroy all unused investigational medicinal product supplies, including empty containers, according to these procedures. If the site cannot meet Gilead Science's requirements for disposal, arrangements will be made between the site and Gilead Sciences or its representative for destruction or return of unused investigational medicinal product supplies.

All drug supplies and associated documentation will be periodically reviewed and verified by the study monitor over the course of the study.

## 9.1.8. Inspections

The investigator should understand that source documents for this trial should be made available to appropriately qualified personnel from Gilead Sciences and its representatives, to IRBs/IECs/ECs, or to regulatory authority or health authority inspectors.

## 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

## 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB/IEC/EC in accordance with local requirements and receive documented approval before modifications can be implemented.

## 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agency. Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

- The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
- The study has been completed at all study sites for at least 2 years

No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).

The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation. The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

## 9.3. Joint Investigator/Sponsor Responsibilities

#### 9.3.1. Payment Reporting

Investigators and their study staff may be asked to provide services performed under this protocol, eg, attendance at Investigator's Meetings. If required under the applicable statutory and regulatory requirements, Gilead will capture and disclose to Federal and State agencies any expenses paid or reimbursed for such services, including any clinical trial payments, meal, travel expenses or reimbursements, consulting fees, and any other transfer of value.

## 9.3.2. Access to Information for Monitoring

In accordance with regulations and guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the eCRF.

The monitor is responsible for routine review of the eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records (including electronic medical records, if applicable) needed to verify the entries on the eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

## 9.3.3. Monitoring and Oversight of Biomarker Specimens

Biomarker research specimens will be tracked in a manner consistent with Good Clinical Practice by a quality-controlled, auditable, and appropriately validated laboratory information management system, to ensure compliance with data confidentiality as well as adherence to authorized use of specimens as specified in this protocol and in the Informed Consent Form.

## 9.3.4. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

## 9.3.5. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority (ies), IRBs, IECs, and ECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

## 10. REFERENCES

- Adachi E, Koibuchi T, Imai K, Kikuchi T, Shimizu S, Koga M, et al. Hemophagocytic syndrome in an acute human immunodeficiency virus infection. Internal medicine (Tokyo, Japan) 2013;52 (5):629-32.
- Akriviadis E, Botla R, Briggs W, Han S, Reynolds T, Shakil O. Pentoxifylline improves short-term survival in severe acute alcoholic hepatitis: a double-blind, placebo-controlled trial. Gastroenterology 2000;119 (6):1637-48.
- Angeli P, Gines P, Wong F, Bernardi M, Boyer TD, Gerbes A, et al. Diagnosis and management of acute kidney injury in patients with cirrhosis: revised consensus recommendations of the International Club of Ascites. Gut 2015;64 (4):531-7.
- Cederbaum AI, Yang L, Wang X, Wu D. CYP2E1 Sensitizes the Liver to LPS- and TNF alpha-Induced Toxicity via Elevated Oxidative and Nitrosative Stress and Activation of ASK-1 and JNK Mitogen-Activated Kinases. International journal of hepatology 2012;2012:582790.
- Chayanupatkul M, Liangpunsakul S. Alcoholic hepatitis: a comprehensive review of pathogenesis and treatment. World J Gastroenterol 2014;20 (20):6279-86.
- European Association for the Study of the Liver (EASL). EASL clinical practical guidelines: management of alcoholic liver disease. J Hepatol 2012;57 (2):399-420.
- Fujino G, Noguchi T, Matsuzawa A, Yamauchi S, Saitoh M, Takeda K, et al. Thioredoxin and TRAF family proteins regulate reactive oxygen species-dependent activation of ASK1 through reciprocal modulation of the N-terminal homophilic interaction of ASK1. Mol Cell Biol 2007;27 (23):8152-63.
- Fujisawa T, Takeda K, Ichijo H. ASK family proteins in stress response and disease. Molecular biotechnology 2007;37 (1):13-8.
- Gao B, Bataller R. Alcoholic liver disease: pathogenesis and new therapeutic targets. Gastroenterology 2011;141 (5):1572-85.
- Gerczuk PZ, Breckenridge DG, Liles JT, Budas GR, Shryock JC, Belardinelli L, et al. An apoptosis signal-regulating kinase 1 inhibitor reduces cardiomyocyte apoptosis and infarct size in a rat ischemia-reperfusion model. J Cardiovasc Pharmacol 2012;60 (3):276-82.
- Hislop WS, Bouchier IA, Allan JG, Brunt PW, Eastwood M, Finlayson ND, et al. Alcoholic liver disease in Scotland and northeastern England: presenting features in 510 patients. Q J Med 1983;52 (206):232-43.

- Imoto K, Kukidome D, Nishikawa T, Matsuhisa T, Sonoda K, Fujisawa K, et al. Impact of mitochondrial reactive oxygen species and apoptosis signal-regulating kinase 1 on insulin signaling. Diabetes 2006;55 (5):1197-204.
- Jinjuvadia R, Liangpunsakul S, Translational R, Evolving Alcoholic Hepatitis Treatment C. Trends in Alcoholic Hepatitis-related Hospitalizations, Financial Burden, and Mortality in the United States. J Clin Gastroenterol 2015;49 (6):506-11.
- Louvet A, Labreuche J, Artru F, Boursier J, Kim DJ, O'Grady J, et al. Combining Data From Liver Disease Scoring Systems Better Predicts Outcomes of Patients With Alcoholic Hepatitis. Gastroenterology 2015;149 (2):398-406 e8.
- Louvet A, Naveau S, Abdelnour M, Ramond MJ, Diaz E, Fartoux L, et al. The Lille model: a new tool for therapeutic strategy in patients with severe alcoholic hepatitis treated with steroids. Hepatology 2007;45 (6):1348-54.
- Louvet A, Wartel F, Castel H, Dharancy S, Hollebecque A, Canva-Delcambre V, et al. Infection in patients with severe alcoholic hepatitis treated with steroids: early response to therapy is the key factor. Gastroenterology 2009;137 (2):541-8.
- Lucey MR, Mathurin P, Morgan TR. Alcoholic hepatitis. N Engl J Med 2009;360 (26):2758-69.
- Mathurin P, O'Grady J, Carithers RL, Phillips M, Louvet A, Mendenhall CL, et al. Corticosteroids improve short-term survival in patients with severe alcoholic hepatitis: meta-analysis of individual patient data. Gut 2011;60 (2):255-60.
- Matsuzawa A, Saegusa K, Noguchi T, Sadamitsu C, Nishitoh H, Nagai S, et al. ROS-dependent activation of the TRAF6-ASK1-p38 pathway is selectively required for TLR4-mediated innate immunity. Nature immunology 2005;6 (6):587-92.
- Meagher EA, Barry OP, Burke A, Lucey MR, Lawson JA, Rokach J, et al. Alcohol-induced generation of lipid peroxidation products in humans. J Clin Invest 1999;104 (6):805-13.
- Michelena J, Altamirano J, Abraldes JG, Affo S, Morales-Ibanez O, Sancho-Bru P, et al. Systemic inflammatory response and serum lipopolysaccharide levels predict multiple organ failure and death in alcoholic hepatitis. Hepatology 2015;62 (3):762-72.
- Mnich SJ, Blanner PM, Hu LG, Shaffer AF, Happa FA, O'Neil S, et al. Critical role for apoptosis signal-regulating kinase 1 in the development of inflammatory K/BxN serum-induced arthritis. Int Immunopharmacol 2010;10 (10):1170-6.
- Nagai H, Noguchi T, Takeda K, Ichijo H. Pathophysiological Roles of ASK1-MAP Kinase Signaling Pathways. Journal of Biochemistry and Molecular Biology 2007;40 (1):1-6.

CONFIDENTIAL Page 94 04 August 2017

- Nakagawa H, Hirata Y, Takeda K, Hayakawa Y, Sato T, Kinoshita H, et al. Apoptosis signal-regulating kinase 1 inhibits hepatocarcinogenesis by controlling the tumor-suppressing function of stress-activated mitogen-activated protein kinase. Hepatology 2011;54 (1):185-95.
- Nakagawa H, Maeda S, Hikiba Y, Ohmae T, Shibata W, Yanai A, et al. Deletion of apoptosis signal-regulating kinase 1 attenuates acetaminophen-induced liver injury by inhibiting c-Jun N-terminal kinase activation. Gastroenterology 2008;135 (4):1311-21.
- Nakamura T, Kataoka K, Fukuda M, Nako H, Tokutomi Y, Dong YF, et al. Critical role of apoptosis signal-regulating kinase 1 in aldosterone/salt-induced cardiac inflammation and fibrosis. Hypertension 2009;54 (3):544-51.
- Nguyen-Khac E, Thevenot T, Piquet MA, Benferhat S, Goria O, Chatelain D, et al. Glucocorticoids plus N-acetylcysteine in severe alcoholic hepatitis. N Engl J Med 2011;365 (19):1781-9.
- Noguchi H, Yamada S, Nabeshima A, Guo X, Tanimoto A, Wang KY, et al. Depletion of apoptosis signal-regulating kinase 1 prevents bile duct ligation-induced necroinflammation and subsequent peribiliary fibrosis. Am J Pathol 2014:1-18.
- O'Shea RS, Dasarathy S, McCullough AJ, Practice Guideline Committee of the American Association for the Study of Liver D, Practice Parameters Committee of the American College of G. Alcoholic liver disease. Hepatology 2010;51 (1):307-28.
- O'Shea RS, McCullough AJ. Treatment of alcoholic hepatitis. Clin Liver Dis 2005;9 (1):103-34.
- Rudler M, Mouri S, Charlotte F, Lebray P, Capocci R, Benosman H, et al. Prognosis of treated severe alcoholic hepatitis in patients with gastrointestinal bleeding. J Hepatol 2015;62 (4):816-21.
- Singal AK, Guturu P, Hmoud B, Kuo YF, Salameh H, Wiesner RH. Evolving frequency and outcomes of liver transplantation based on etiology of liver disease.

  Transplantation 2013;95 (5):755-60.
- Spahr L, Rubbia-Brandt L, Frossard JL, Giostra E, Rougemont AL, Pugin J, et al. Combination of steroids with infliximab or placebo in severe alcoholic hepatitis: a randomized controlled pilot study. J Hepatol 2002;37 (4):448-55.
- Taieb J, Mathurin P, Elbim C, Cluzel P, Arce-Vicioso M, Bernard B, et al. Blood neutrophil functions and cytokine release in severe alcoholic hepatitis: effect of corticosteroids. J Hepatol 2000;32 (4):579-86.
- Takeda K, Noguchi T, Naguro I, Ichijo H. Apoptosis signal-regulating kinase 1 in stress and immune response. Annu Rev Pharmacol Toxicol 2008;48:199-225.

CONFIDENTIAL Page 95 04 August 2017

- Terada Y, Inoshita S, Kuwana H, Kobayashi T, Okado T, Ichijo H, et al. Important role of apoptosis signal-regulating kinase 1 in ischemic acute kidney injury. Biochem Biophys Res Commun 2007;364 (4):1043-9.
- Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, et al. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med 2015;372 (17):1619-28.
- Tobiume K, Matsuzawa A, Takahashi T, Nishitoh H, Morita K, Takeda K, et al. ASK1 is required for sustained activations of JNK/p38 MAP kinases and apoptosis. EMBO reports 2001;2 (3):222-8.
- Tobiume K, Saitoh M, Ichijo H. Activation of apoptosis signal-regulating kinase 1 by the stress-induced activating phosphorylation of pre-formed oligomer. Journal of cellular physiology 2002;191 (1):95-104.
- Toldo S, Breckenridge DG, Mezzaroma E, Tassell BW, Shryock J, Kannan H, et al. Inhibition of apoptosis signal-regulating kinase 1 reduces myocardial ischemia-reperfusion injury in the mouse. Journal of the American Heart Association 2012;1 (5):e002360.
- Watanabe T, Otsu K, Takeda T, Yamaguchi O, Hikoso S, Kashiwase K, et al. Apoptosis signal-regulating kinase 1 is involved not only in apoptosis but also in non-apoptotic cardiomyocyte death. Biochem Biophys Res Commun 2005;333 (2):562-7.
- Xie Y, Ramachandran A, Breckenridge DG, Liles JT, Lebofsky M, Farhood A, et al. Inhibitor of apoptosis signal-regulating kinase 1 protects against acetaminophen-induced liver injury. Toxicol Appl Pharmacol 2015;286 (1):1-9.
- Yokoi T, Fukuo K, Yasuda O, Hotta M, Miyazaki J, Takemura Y, et al. Apoptosis signal-regulating kinase 1 mediates cellular senescence induced by high glucose in endothelial cells. Diabetes 2006;55 (6):1660-5.
- Zhang R, Al-Lamki R, Bai L, Streb JW, Miano JM, Bradley J, et al. Thioredoxin-2 inhibits mitochondria-located ASK1-mediated apoptosis in a JNK-independent manner. Circ Res 2004;94 (11):1483-91.
- Ziol M, Tepper M, Lohez M, Arcangeli G, Ganne N, Christidis C, et al. Clinical and biological relevance of hepatocyte apoptosis in alcoholic hepatitis. J Hepatol 2001;34 (2):254-60.

## 11. APPENDICES

| Appendix 1. | Investigator Signature Page |
|-------------|-----------------------------|
| Appendix 2. | Study Procedures Table |

Appendix 3. Pregnancy Precautions, Definition for Female of Childbearing Potential, and

Contraceptive Requirements

Appendix 4. Child-Pugh-Turcotte (CPT) Classification of the severity of cirrhosis

## Appendix 1. Investigator Signature Page

## GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404

## STUDY ACKNOWLEDGEMENT

A Phase 2, Double-Blind, Randomized Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 in Combination with Prednisolone versus Prednisolone Alone in Subjects with Severe Alcoholic Hepatitis (AH)

## GS-US-416-2124, Amendment 3, 04 August 2017

| OS-OS-410-2124, Amenun | ient 5, 04 August 2017 |
|---|---|
| This protocol has been approved by Gilead Science this approval. | es, Inc. The following signature documents |
| Chuhar Chung, MD Medical Monitor | o.g |
| Date 4 August 2017 | |
| INVESTIGATOR | STATEMENT |
| I have read the protocol, including all appendices, a details for me and my staff to conduct this study as outlined herein and will make a reasonable effort to designated. | described. I will conduct this study as |
| I will provide all study personnel under my supervi<br>information provided by Gilead Sciences, Inc. I wil<br>that they are fully informed about the drugs and the | l discuss this material with them to ensure |
| Principal Investigator Name (Printed) | Signature |
| Date | Site Number |

## Appendix 2. Study Procedures Table

| | Scree | reening <sup>a</sup> Treatment <sup>b</sup> Post-Treatment | | | | | | | | | | | | | | Unscheduled<br>Visit | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | eline/ | | eek<br>1 | V | Veek<br>2 | 78.0 | eek<br>3 | | eek 4/<br>CoT <sup>t</sup> | Week<br>6 | Week<br>8 u | Week<br>12 <sup>u</sup> | Week<br>16 | Week<br>20 | Week<br>24 <sup>u</sup> | Follow Up<br>visit v |
| | -14 d | lays | 200 | ay 1 | | ±3 days | | | | | | | | | | ±5 days | | | | | | |
| Informed Consent | Х | | | | | | | | | | | | | | | | | | | | | |
| Review Inclusion/Exclusion<br>Criteria | X | | - 5 | X | | X | | | | | | | | | | | | | | | | |
| Medical History | X | 2 | Î | | 35 | | | | | | | | 8 | | 3 | 3 | | 8 | | | | |
| AUDIT / SADQ <sup>c</sup> | Х | | | | | | | | | | | | | | | | | | | | | |
| QoL (CLDQ) c | | | 2 | X | 82 | | | | | | | X | 6 85 | | | | | X | , | | | |
| Alcohol Consumption | Х | ş | 1 8 | X | | X | 3 | X | | X | | X | X | X | X | X | X | X | | | | |
| Complete Physical Exam <sup>d</sup> | X | 9 | . 9 | X | | X | | X | 1 | X | | X | X | X | X | X | X | X | | | | |
| Height | X | | | | | | 3 | | 9 | | | | 6 | | 3 | . 3 | | 55 | | | | |
| Weight | X | \$ | 8 | X | 5. | | 3 | | | | | X | 8 | | X | | | X | 8 | | | |
| Vital Signs | X | Q. | X | | X | | X | | X | | X | | X | X | X | X | X | X | | | | |
| 12-lead ECG <sup>e</sup> | Х | | X | | 5 | | | | | X | | | X | | | | 23 | | | | | |
| | Local lab | Central lab | Local lab | Central lab | Local lab | Central lab | Local lab | Central lab | Local lab | Central lab | Local lab | Central lab | | | | | | | | | | |
| Urine Drug Screen <sup>f</sup> | X | X | | | 8. | | | | | S. | | es. | 35 | | | | | 50 | | | | |
| Urinalysis <sup>g</sup> | Х | | | 8 | | 13 | | | | 8 | | | E 55 | | | . 3 | | 54 | | | | |
| HRSe | X | | 2 | X | | X | 9 | X | | X | | X | X | X | X | x | X | X | X | Х | | |
| Infection <sup>e</sup> | X | | | X | | X | | X | | X | | X | х | X | X | X | X | X | X | X | | |
| Hematology | X | X | 8 | Х | 8 | X | 3 8 | X | | X | | X | X | X | X | X | X | X | X | X | | |
| Chemistry <sup>i</sup> | X | X | Х | X | X | X | Х | X | X | X | X | X | X | X | X | X | X | X | X | Х | | |

| | Scre | ening <sup>a</sup> | | Treatment <sup>b</sup> | | | | | | | | | | | | Unscheduled<br>Visit | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | D- | seline/ | V | Veek<br>1 | V | Veek<br>2 | V | Veek<br>3 | | eek 4/<br>CoT <sup>t</sup> | Week<br>6 | Week<br>8" | Week<br>12 <sup>u</sup> | Week<br>16 | Week<br>20 | Week<br>24 <sup>u</sup> | Follow Up<br>visit v | |
| | -14 | days | | ay 1 | - Ct | | | | ±3 d | ays | | | 7 | | | | ±5 days | | - | |
| Hepatitis B and C, HIV | X | X | | | | | | | | | | | | | | | | | | |
| Coagulation Tests <sup>k</sup> | X | X | X | X | 165 | X | | X | | X | | X | x | X | X | X | X | X | X | X |
| Pregnancy Test <sup>1</sup> | X<br>(urine) | X<br>(serum) | ) | Х | | | | | | | | Х | | X | X | X | х | X | | |
| | Local Lab | Central Lab | Local Lab | Central Lab | Local Lab | Central Lab | Local Lab | Central Lab | Local Lab | Central Lab | Local Lab | Central Lab | | | | | | | | |
| Blood Cultures | X | | | | 16 | | | | | | | | | | | | | 23 | | |
| Ascitic Fluid Tap <sup>m</sup> | X | | | | | | | | | | | | | | | | | | | |
| Liver Biopsy | Xn | | | | | | | | | | | | | | | | | 5) | | A A |
| Insulin | | X | | X | | | | | | | | X | | | X | | | X | | |
| Lipid Profile | | X | | X | | | | | | | | X | | | X | | | X | | |
| Blood Sample for<br>Biomarkers° | | X | 5 | X | 8 | X | 30 - 30 | X | | 10 | | X | | X | X | | | X | | 9 |
| Urine Sample for Biomarkers | | | r. | X | 88<br>(15 | 10 | | | | | | X | | | | j | | X | 8 | |
| ELF test, LOXL2 | | | | X | | | | | | | | X | | | X | | | X | | |
| Hemoglobin A1c | | | | X | | | | | | | | | | | X | | | X | | |
| Hepatic Encephalopathy | | x | | | | x | | X | | X | | X | X | X | X | X | X | X | X | X |
| Ascites <sup>d</sup> | 7 | Xh | 45 | | | X | | X | | X | | X | X | X | X | X | X | X | X | X |
| Chest X-ray | | X | e<br>v | | - Q | | × | | 9 | | | | | | | × | | | | |
| Liver Ultrasound | | X | 2 | | 3 | | | | 6 | | | | | | | | | | | |
| Review Concomitant<br>Medications | | X | ð | X | | X | | X | | X | | X | X | Х | X | X | X | X | X | Х |

| | Screening <sup>a</sup> | | | Treatment <sup>b</sup> | | | | | | Unscheduled<br>Visit | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline/ - | Week<br>1 | Week<br>2 | Week<br>3 | Week 4/<br>EoT <sup>t</sup> | Week<br>6 | Week<br>8 u | Week<br>12 <sup>u</sup> | Week<br>16 | Week<br>20 | Week<br>24 <sup>u</sup> | Follow Up<br>visit v | Ē |
| | -14 days | Day 1 | | | ±3 days | | | | | | ±5 days | | - 6: | |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Sparse PK Sample <sup>p</sup> | | X | X | X | | $X^p$ | | | | | | | | |
| Stool Collection | | X | | | | X | | | | | | X | | |
| Randomization <sup>q</sup> | | X | | | | | | | | | | | | |
| GS-4997 Dispensing | | X | | | | | | | | | 6.<br>E | | | |
| Prednisolone Dispensing | | X | X | | X | 3. | | | | | 6 | | | |
| PPD | | | | | | | | | | | | | | |
| Genomic Sample <sup>s</sup> | | X | | | | | | | | | | | | |
| Study Drug Adherence | | | X | X | X | X | | | | | | | | |
| FibroScan <sup>w</sup> | | X | | | | X | | | | | 8 | X | | |
| Lille Score <sup>x</sup> | | | X | X | X | X | | | | | | | | |

- The visit window may be extended under special circumstances with explicit approval of the Medical Monitor. Subjects who fail to meet eligibility criteria due to an abnormal laboratory result may undergo re-testing of the abnormal analyte once during the Screening window. This will be done at the discretion of the investigator and also with prior approval of the Medical Monitor. The following laboratory tests will be collected at Screening for testing at both the local and central laboratories: urine drug screen, hematology, chemistry, and coagulation tests. Eligibility will be based on local laboratory results. For urine drug screen, local laboratory testing done within 10 days of the Screening visit may be used to determine eligibility. For hepatitis B serology, hepatitis C serology, and HIV serology, these tests will be sent to both the local and central laboratories with eligibility based on local laboratory testing. A urine pregnancy test will also be done at Screening but only sent to the local laboratory and be the basis for eligibility. A serum pregnancy test will be sent only to the central laboratory at Screening.
- b During the hospitalization period, subjects will be evaluated daily with assessments to include a review of adverse events, concomitant medications, study drug adherence, and a symptom-directed PE including assessments for ascites and HE. Findings based on these assessments and laboratory investigations obtained by treating physicians as part of routine care will be assessed by the investigator for triggers that may necessitate further evaluation and/or treatment discontinuation and managed accordingly per Section 7 of the protocol.
- c A Legally Authorized Representative may assist the subject in completing the questionnaires. If the subject is unable or refuses to complete a questionnaire, this should be documented on the relevant eCRF.
- d Perform a complete Physical Exam with a focus on ascites and encephalopathy.
- e Please see Section 6.9 for description of assessments and record diagnosis/abnormal findings as an AE.
- f Drug screen for amphetamines, cocaine and opiates (ie heroin, morphine).

- g Urinalysis (routine and microscopic) and culture to be performed by local lab.
- Subjects with evidence of sepsis or gastrointestinal bleeding may be treated for a minimum of 2 days with appropriate antibiotics. Once deemed stable, subject may continue Screening and randomized if eligible.
- i Chemistry will include: alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin, alkaline phosphatase, bicarbonate, blood urea nitrogen, calcium, chloride, creatinine, glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, gamma-glutamyl transferase (GGT). Chemistry must be collected for both local and central lab at Baseline/Day1, Week 1, Week 2, Week 3, and Week 4 for Lille Score
- j Local laboratory results for Hepatitis B and C and HIV Serology done within 10 days of the Screening visit may be used to determine eligibility.
- k Coagulation Panel includes: PT, PTT and INR. Coagulation must be collected for both local and central lab at Baseline/Day visit for Lille Score.
- 1 Females of childbearing potential only. Serum pregnancy test at Screening done at central lab. Urine pregnancy test at Screening and other visits.
- m Paracentesis with ascitic fluid cell count, differential, and culture will be performed if clinically-detectable ascites is present.
- Liver biopsy obtained during the current hospital admission prior to Screening is acceptable. Liver biopsy can be performed up to 7 days post Baseline/Day 1. However, if biopsy results are not consistent with AH, the subject will discontinue study drug within 3 days of receipt of liver biopsy result, attend an EoT visit as soon as possible and attend a 30-day FU visits and be withdrawn from the study. If the liver biopsy sample is inadequate for a pathologic diagnosis of AH, but does not reveal an alternative etiology, the subject may remain in the study.
- o Blood for Biomarkers collection will occur at all study sites. Biomarker phospho-p38 blood sample will be collected prior to the first dose of study drug only at US study sites.
- p Please refer to Section 6.4.1 for sample collection instructions. If subject's last dose of study drug is prior to the Week 4 visit, PK sample can still be collected at Week 4 as long as last dose date and time is prior to sample collection. If a subject requires hemodialysis/ hemoperfusion/peritoneal dialysis therapy, please refer to Section 6.4.1 for collection instructions.
- q Stratification of MELD < or ≥ 25 at Screening will be based on local laboratory testing and utilize the following calculator: http://www.mdcalc.com/original-meld-score-pre-2016-model-for-end-stage-liver-disease</p>
- r PPD
- s PPU
- t Subjects discontinuing treatment at any time prior to Week 4 for any reason should complete the procedures required for the Week 4 / End of Treatment Visit. These subjects will require a phone contact between study days 28-35 to assess for mortality and liver transplantation and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study.
- u Subjects with a Week 8, Week 12, or Week 24 visit prior to Day 56, Day 84, or Day 168 respectively will be required to have a telephone contact between Days 56-63, Days 84-89, or 168-173 respectively to assess for mortality and liver transplantation.
- v Subjects whose liver biopsy results are not consistent with AH or whose HIV or hepatitis B or C serologies from the central laboratory are positive, must stop study drug within 3 days of receipt of results. Subjects whose serum pregnancy testing from the central laboratory is positive at Screening must stop study drug immediately upon receipt of this result. All subjects stopping study drug for these reasons should attend an EoT visit as soon as possible and have a follow up visit 30 days after their last dose of study drug, prior to being withdrawn from the study. If the liver biopsy sample is inadequate for a pathologic diagnosis of AH, but does not reveal an alternative etiology, the subject may remain in the study.
- w At sites where available and only on subjects without ascites.
- x Sites to calculate based on local laboratory results using the following calculator: http://www.mdcalc.com/lille-model-alcoholic-hepatitis/. When using the calculator, ensure the Day 7 total bilirubin is changed to Weeks 2, 3, and 4 values at the appropriate time points.

# Appendix 3. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

## 1) Definitions

## a. Definition of Childbearing Potential

For the purposes of this study, a female born subject is considered of childbearing potential following the initiation of puberty (Tanner stage 2) until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure.

Women are considered to be in a postmenopausal state when they are  $\geq 54$  years of age with cessation of previously occurring menses for  $\geq 12$  months without an alternative cause.

Permanent sterilization includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age.

## b. Definition of Male Fertility

For the purposes of this study, a male born subject is considered fertile after the initiation of puberty unless permanently sterile by bilateral orchidectomy or has medical documentation of permanent male infertility.

## 2) Contraception Requirements for Female Subjects

## a. Study Drug Effects on Pregnancy and Hormonal Contraception

GS-4997 is contraindicated in pregnancy as a malformation effect is suspected, based on non-clinical data. In rats and rabbits, GS-4997 administration was associated with effects on embryo-fetal development at maternally toxic doses. This included total litter loss, increased resorptions and post implantation loss, reduced fetal weights, and visceral and skeletal malformations and variations. Embryofetal effects were observed in rats and rabbits at exposures (AUC24hr) that were 62- and 12-fold higher, respectively, than the GS-4997 steady state exposure in NASH subjects at the maximum human dose of 18 mg once daily. The NOELs for embryofetal development in rats and rabbits were 15 and 10 mg/kg/day, respectively. The exposure margins at these doses as compared to the maximum proposed human dose are 12 - and 3-fold, respectively.

Preclinical data indicate that GS-4997 is unlikely to reduce the exposure of hormonal contraceptives through induction of human drug metabolizing enzymes or drug transporters. This is supported by clinical DDI data, which demonstrated multiple doses of GS-4997 did not result in increased activity of CYP3A4 or P-gp based on plasma exposures of sensitive probe substrates (midazolam and digoxin). Similarly, preclinical and clinical data indicate GS-4997 is unlikely to cause a clinically relevant increase in the exposure of hormonal contraceptives through inhibition of drug metabolizing enzymes or drug transporters. Please refer to the latest version of the investigator's brochure for additional information.

## b. Contraception Requirements for Female Subjects of Childbearing Potential

The inclusion of female subjects of childbearing potential requires the use of highly effective contraceptive measures. They must have a negative serum pregnancy test at Screening and a negative pregnancy test on the Baseline/Day 1 visit prior to randomization. Pregnancy tests will be performed at monthly intervals thereafter. Female subjects must agree to one of the following from Screening until 90 days after the last dose of study drug.

• Complete abstinence from intercourse of reproductive potential. Abstinence is an acceptable method of contraception only when it is in line with the subject's preferred and usual lifestyle.

Or

- Consistent and correct use of 1 of the following methods of birth control listed below.
  - Intrauterine device (IUD) with a failure rate of < 1% per year
  - Tubal sterilization
  - Essure micro-insert system (provided confirmation of success 3 months after procedure)
  - Vasectomy in the male partner (provided that the partner is the sole sexual partner and had confirmation of surgical success 3 months after procedure)
- The above described methods are considered preferred methods of highly effective contraception in this protocol.
  - Should female subjects wish to use a hormonally based method, use of a male condom by the female subject's male partner is required. Subjects who utilize a hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing. Hormonally-based contraceptives permitted for use in this protocol are as follows:
    - Hormonal methods (each method *must* be used with a condom in the male partner)
      - Oral contraceptives (either combined or progesterone only)
      - Injectable progesterone
      - Implants of levonorgestrel
      - Transdermal contraceptive patch
      - Contraceptive vaginal ring

Female subjects must also refrain from egg donation and in vitro fertilization during treatment and until at least 90 days after the last dose of study drug.

## 3) Contraception Requirements for Male Subjects

It is theoretically possible that a relevant systemic concentration may be achieved in a female partner from exposure of the male subject's seminal fluid. Therefore, male subjects with female partners of childbearing potential must use condoms during treatment until 90 days after the last dose of study drug. Female partners of male study subjects should consider using one of the above methods of contraception as well.

Male subjects must also refrain from sperm donation during treatment and until at least 90 days after the last dose of study drug.

## 4) Unacceptable Birth Control Methods

Birth control methods that are unacceptable include periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM). Female condom and male condom should not be used together.

## 5) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study, or if they become pregnant within 90 days of last study drug dose. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant during the study must report the information to the investigator. Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.6.2.1.

## Appendix 4. Child-Pugh-Turcotte (CPT) Classification of the severity of cirrhosis

| | POINTS | | |
|---|---|---|---|
| | 1 | 2 | 3 |
| Encephalopathy | None | Grade 1-2 (medication-controlled) | Grade 3-4 (medication-refractory) |
| Ascites | None | Mild/Moderate<br>(diuretic-responsive) | Severe (diuretic-refractory) |
| Bilirubin (mg/dL) | < 2 | 2-3 | > 3 |
| Albumin (g/dL) | > 3.5 | 2.8-3.5 | < 2.8 |
| INR | < 1.7 | 1.7-2.3 | > 2.3 |

Note: if the either ascites or encephalopathy is "none" because the patient is taking medication which has controlled the symptoms, the scoring should be 2 points (not 1 point).

CPT score is obtained by adding the points for each parameter

CPT class is scored as: A = 5-6 points

B = 7-9 points

C = 10-15 points